# Johnson & Johnson Vision Care, Inc.

# Clinical Study Protocol

Evaluation of A Marketed Silicone Hydrogel Spherical Lens Used for Monovision Correction of Presbyopia

Protocol CR-6349

Version: 5.0 Amendment 4

Date: 03 September 2019

Investigational Products: ACUVUE® OASYS with Transitions<sup>TM</sup>

Key Words: Presbyopia, Monovision, senofilcon A, Daily Wear, Reusable, Dispensing

## Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155,<sup>1</sup> the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP),<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements.

## **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

## PROTOCOL TITLE, NUMBER, VERSION......6 SPONSOR NAME AND ADDRESS......6 AUTHORIZED SIGNATURES.......7 CHANGE HISTORY 8 COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS ...... 14 1.1. 1.2. 1.3. 1.4. 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES ...... 16 2.1. 2.2. 2.3. 3.1. General Characteristics 17 3.2. 3.3. Exclusion Criteria 18 3.4.

TABLE OF CONTENTS

4.1.

4.2.

4.3.

5.1.

5.2.5.3.

| | 6.1. | Identity of Test Articles | 21 |
|---|---|---|---|
| | 6.2. | Ancillary Supplies/Products | 21 |
| | 6.3. | Administration of Test Articles | 22 |
| | 6.4. | Packaging and Labeling | 22 |
| | 6.5. | Storage Conditions | 22 |
| | 6.6. | Collection and Storage of Samples | 23 |
| | 6.7. | Accountability of Test Articles | 23 |
| 7 | . ST | UDY EVALUATIONS | 24 |
| | 7.1. | Time and Event Schedule | 24 |
| | 7.2. | Detailed Study Procedures | 26 |
| | VIS | SIT 1 | 26 |
| | VIS | SIT 2 | 32 |
| | VIS | SIT 3 | 35 |
| | VIS | SIT 4 | 39 |
| | FIN | NAL EVALUATION | 41 |
| | 7.3. | Unscheduled Visits | 42 |
| | 7.4. | Laboratory Procedures | 44 |
| 8 | S. SU | BJECTS COMPLETION/WITHDRAWAL | |
| | 8.1. | Completion Criteria | 44 |
| | 8.2. | Withdrawal/Discontinuation from the Study | 44 |
| 9 | PR | E-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 45 |
| 1 | 0. D | DEVIATIONS FROM THE PROTOCOL | 45 |
| 1 | 1. S | TUDY TERMINATION | 45 |
| 1 | 2. P | ROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 46 |
| 1 | 3. A | ADVERSE EVENTS | 47 |
| | 13.1. | Definitions and Classifications | 47 |
| | 13.2. | Assessing Adverse Events | 49 |
| | 13. | 2.1. Causality Assessment | 49 |
| | 13. | 2.2. Severity Assessment | 50 |
| | 13.3. | Documentation and Follow-Up of Adverse Events | 50 |
| | 13.4. | Reporting Adverse Events | 51 |
| | 13. | 4.1. Reporting Adverse Events to Sponsor | 52 |
| | | 4.2. Reporting Adverse Events to the Responsible IEC/IRB and I thorities | |
| | 13. | 4.3. Event of Special Interest | 53 |

| 13.5 | 5. | Reporting of Pregnancy | . 53 |
|---|---|---|---|
| 14. | STA | ATISTICAL METHODS | . 53 |
| 14. | 1. | General Considerations. | . 53 |
| 14.2 | 2. | Sample Size Justification | . 53 |
| 14.3 | 3. | Analysis Populations | . 54 |
| 14.4 | 4. | Level of Statistical Significance | . 54 |
| 14.5 | 5. | Primary Analysis | . 54 |
| 14.6 | 5. | Secondary Analysis | . 56 |
| 14. | 7. | Other Exploratory Analyses | . 56 |
| 14.8 | 8. | Interim Analysis | . 56 |
| 14.9 | 9. | Procedure for Handling Missing Data and Drop-Outs | . 56 |
| 14. | 10. | Procedure for Reporting Deviations from Statistical Plan | . 56 |
| 15. | DA | TA HANDLING AND RECORD KEEPING/ARCHIVING | . 56 |
| 15. | 1. | Electronic Case Report Form/Data Collection | . 56 |
| 15.2 | 2. | Subject Record | . 57 |
| 16. | DA | TA MANAGEMENT | . 57 |
| 16. | 1. | Access to Source Data/Document | . 57 |
| 16.2 | 2. | Confidentiality of Information | . 58 |
| 16.3 | 3. | Data Quality Assurance | . 58 |
| 17. | MO | NITORING | . 58 |
| 18. | ETH | HICAL AND REGULATORY ASPECTS | . 59 |
| 18. | 1. | Study-Specific Design Considerations | . 59 |
| 18.2 | 2. | Investigator Responsibility | . 59 |
| 18.3 | 3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | . 59 |
| 18.4 | 4. | Informed Consent | 60 |
| 18.5 | 5. | Privacy of Personal Data | 61 |
| 19. | STU | JDY RECORD RETENTION | 62 |
| 20. | FIN | ANCIAL CONSIDERATIONS | 62 |
| 21. | PUE | BLICATION | 63 |
| 22. | REF | FERENCES | 64 |
| | | X A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | |
| | | X B: PATIENT INSTRUCTION GUIDE | |
| APPE | NDE | X C: PACKAGE INSERT (APPROVED PRODUCT) | . 93 |
| APPE | NDL | X D: BINOCULAR OVER REFRACTION | 122 |

| APPENDIX E: PRESBYOPIC SYMPTOMS QUESTIONNAIRE | 123 |
|-----------------------------------------------------|--------|
| APPENDIX F: OCULAR DOMINANCE | 124 |
| APPENDIX G: AST SENTIO CONTRAST SENSITIVITY TESTING | 125 |
| APPENDIX H: | 132 |
| LIMBAL AND CONJUNCTIVAL (BULBAR) REDNESS | |
| EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING | |
| DETERMINATION OF NEAR ADDITION | 146 |
| NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDU | RE 154 |
| LENS FITTING CHARACTERISTICS | 157 |
| SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS | 164 |
| DETERMINATION OF DISTANCE SPHEROCYLINDRICAL | |
| REFRACTIONS | |
| KERATOMETRY PROCEDURE | |
| DISTANCE AND NEAR VISUAL ACUITY EVALUATION | |
| DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PRO | |
| VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINA | |
| TESTING | |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 196 |
| TABLE OF CONTENTS | |
| Figure 1: Study Flowchart | 13 |
| TABLE OF CONTENTS | |
| Table 1: Test Articles | |
| Table 2: Ancillary Supplies | |
| Table 3: Time and Events | |

## PROTOCOL TITLE, NUMBER, VERSION

Title: Evaluation of A Marketed Silicone Hydrogel Spherical Lens Used for Monovision

Correction of Presbyopia Protocol Number: CR-6349 Version: 5.0 Amendment 4 Date: 03 September 2019

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### MEDICAL MONITOR

Name: Thomas R. Karkkainen, OD, MS, FAAO

Title: Sr. Principal Research Optometrist

Address: 7500 Centurion Parkway, Jacksonville, Florida 32256

Email: TKarkkai@its.jnj.com

The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### **AUTHORIZED SIGNATURES**

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations,<sup>4</sup> ICH guidelines,<sup>2</sup> ISO 14155,<sup>1</sup> and the Declaration of Helsinki.<sup>3</sup>

| Author | See Electronic Signature Report Thomas R. Karkkainen, OD, MS, FAAO Sr. Principal Research Optometrist, Clinical Sciences | DATE |
|---|---|---|
| Clinical Operations<br>Manager | See Electronic Signature Report | DATE |
| Biostatistician | See Electronic Signature Report | DATE |
| Data Management | See Electronic Signature Report | DATE |
| Reviewer | See Electronic Signature Report | DATE |
| Approver | See Electronic Signature Report | DATE |

## **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section | Date |
|---|---|---|---|
| | | Number(s) Affected | |
| 1.0 | Tom | Original Protocol | 25 June 2019 |
| | Karkkainen | | |
| 2.0 | | <ul> <li>Revised the order of Exclusion</li> </ul> | 02 July 2019 |
| Amendment 1 | 32 24 | in both the Synopsis and | |
| | | Section 3.2 Exclusion Criteria. | |
| | | <ul> <li>Revised the order of steps 3.11</li> </ul> | |
| | | and 3.12 in Section 7.2 Detailed | |
| | | Study Procedures to be | |
| | | consistent with the other visits. | |
| | | <ul> <li>Updated the Version and Date</li> </ul> | |
| | | throughout the Protocol. | |
| 3.0 | Tom | <ul> <li>Title page, synopsis and</li> </ul> | 26 July 2019 |
| Amendment 2 | Karkkainen | flowchart- removed references | |
| | | to randomization. | |
| | | <ul> <li>Section 2.1-corrected grammar</li> </ul> | |
| | | my removing the word "how". | |
| 4.0 | Tom | <ul> <li>Section 7.2 visit 3 instructions</li> </ul> | 08 August |
| Amendment 3 | Karkkainen | corrected to state subjects must | 2019 |
| | | attend visit 3 with their habitual | |
| | | contact lenses and also removed | |
| | | "if applicable" after lens | |
| | | removal. | |
| 5.0 | Tom | <ul> <li>Revised Section 11.0 Study</li> </ul> | 03 September |
| Amendment 4 | Karkkainen | Termination | 2019 |
| | | <ul> <li>Updated Sections 14.2 Sample</li> </ul> | |
| | | Size Justification, 14.5 Primary | |
| | | Analysis, and 14.6 Secondary | |
| | | Analysis | |
| | | <ul> <li>Updated the Version and Date</li> </ul> | |
| | | throughout the Protocol. | |

# **SYNOPSIS**

| Protocol Title | Evaluation of A Marketed Silicone Hydrogel Spherical Lens<br>Used for Monovision Correction of Presbyopia |
|---|---|
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Development Phase, Phase 2 |
| Trial Registration | This study will be registered on ClinicalTrials.gov. |
| Test Article(s) | Investigational Product: Over-labeled ACUVUE® OASYS with Transitions <sup>TM</sup> |
| Wear and Replacement<br>Schedules | Wear Schedule: The lenses will be used on a daily reusable basis. |
| | Replacement Schedule: The lenses will be worn for approximately 2 weeks. A new set of lenses will be given to the subject at Visit 3 and the lenses will also be replaced if lost or damaged. |
| Objectives | This study is an evaluation of the visual performance and subjective responses of ACUVUE® OASYS with Transitions <sup>TM</sup> fit as monovision. |
| Study Endpoints | Primary endpoints: logMAR visual acuity scores, and CLUE vision scores |
| | Other endpoints: qCSF (Site 1036 only) |
| Study Design | This is a single-masked, dispensing clinical trial. A total of approximately 48 myopic and 32 hyperopic eligible subjects will be targeted to complete the study. At Visit 1, the subjects will be fit in the study lens, optimized if required and wear the study lenses for approximately 2 weeks. |
| | At Visit 2, the endpoints will be measured, and the subjects will be scheduled for Visit 3 after a 7±3 day wash-out. |
| | The subjects will return to Visit 3 and complete a baseline and be fit with the same lens power that was dispensed at Visit 1 (No Optimizations). |
| | The subjects will return for Visit 4 after wearing the final lens pair for approximately 2 weeks. The endpoint measurements will be repeated, and the final evaluation completed. |
| | The primary endpoints will be visual performance scores and |

| | the CLUE vision scores. |
|---|---|
| | See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations. |
| Sample Size | A total of approximately 80 will be targeted to complete. |
| Study Duration | The study will last approximately 3 to 5 months. |
| Anticipated Study Population Healthy male and female volunteers with presbyop screened as per criteria outlined below. All volunt have baseline measurements taken to ensure eligible baseline procedures will occur after informed consobtained. Subjects will have medical and contact I recorded, baseline questionnaires completed, and read anterior segment status determined. | |
| Eligibility Criteria | <ul> <li>Potential subjects must satisfy all of the following criteria to be enrolled in the study</li> <li>Inclusion Criteria after Screening</li> <li>1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.</li> <li>2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.</li> <li>3. The subject must be between 40 and 70 years of age at the time of screening.</li> <li>4. Subjects must own a wearable pair of spectacles if required for their distance vision.</li> <li>5. The subject must be an adapted monovision soft contact lens wearer in both eyes (i.e., worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month of more duration).</li> <li>Inclusion Criteria after Baseline</li> <li>6. The subject's distance spherical equivalent refraction must be in the range of +3.50 D to -4.00 D in each eye.</li> <li>7. The subject's refractive cylinder must be ≤1.00 D in each eye.</li> <li>8. The subject's ADD power must be in the range of +0.75 D to +2.50 D.</li> <li>9. The subject must have best corrected distance visual acuity of 20/20<sup>-3</sup> or better in each eye.</li> <li>Potential subjects who meet any of the following criteria will</li> </ul> |
| | Potential subjects who meet any of the following criteria will |

be excluded from participating in the study:

Exclusion Criteria after Screening

- 1. Currently Pregnant or lactating.
- 2. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g., hepatitis, tuberculosis).
- 3. Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g., Accutane), oral tetracyclines, oral phenothiazines (e.g., Haldol, Mellaril, Thorazine, Elavil, Pamelor, Compazine), systemic steroids.
- 4. Any previous, or planned, ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, dacryocystorhinostomy, etc.).
- 5. Use of any ocular medication, with the exception of rewetting drops.
- 6. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
- 7. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
- 8. Any known hypersensitivity or allergic reaction to OPTI-FREE® Puremoist® care cleaning solution, non-preserved rewetting drop solution or sodium fluorescein.
- 9. History of herpetic keratitis.
- 10. Entropion, ectropion, chalazia, glaucoma, history of recurrent corneal erosions.
- 11. A history of amblyopia, strabismus or binocular vision abnormality.

## Exclusion Criteria after Baseline

- 12. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
- 13. Any ocular infection or inflammation.
- 14. Any ocular abnormality that may interfere with contact

| | lens wear. |
|---|---|
| | 15. Any active or ongoing ocular or systemic allergies that |
| | may interfere with contact lens wear. |
| Disallowed | Concomitant medications will be documented during |
| Medications/Interventions | screening and updated during the study. Disallowed |
| | medications and therapies are medications or therapies that |
| | contraindicate contact lens wear. See the Exclusion criteria |
| | for specific details. |
| Measurements and | logMAR Visual acuity, Subjective responses for vision using |
| Procedures | the CLUE questionnaire, qCSF (Site 1036 only). |
| Microbiology or Other | None |
| Laboratory Testing | |
| Study Termination | The occurrence of one or more Unanticipated Adverse Device |
| | Effect (UADE), or any SAE where relationship to study agent |
| | cannot be ruled out, will result in stopping further dispensing |
| | investigational product. In the event of a UADE or SAE, the |
| | Sponsor Medical Monitor may unmask the treatment regimen |
| | of subject(s) and may discuss this with the Principal |
| | Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study- | OPTI-FREE® Puremoist® multi-purpose care solution, |
| Specific Materials | Rewetting drops, lens cases, glass vials, saline, ETDRS light |
| | cabinet, logMAR charts, and Near logMAR charts. |
| Principal Investigator(s) | A full list of Principal Investigators, clinical sites, and |
| and Study | institutions is kept separately from the Study Protocol and is |
| Institution(s)/Site(s) | included in the study Trial Master File. |
| | I |

Figure 1: Study Flowchart



#### COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required For Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience

BCC Binocular Crossed Cylinder BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations

CLDEQ-8 Contact Lens Dry Eye Questionnaire-8

CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus

IB Investigator's Brochure ICF Informed Consent Form

ICH International Council for Harmonization
IDE Investigational Device Exemption
IEC Independent Ethics Committee
IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision, Inc.

LC Limbus Center

LogMAR Logarithm of Minimal Angle of Resolution

LSM Least Square Means

MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections

OHSR Office for Human Subjects Research

OS Left Eye OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator
PIG Patient Instruction Guide
PQC Product Quality Complaint
PRO Patient Reported Outcome

QA Quality Assurance QC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

Johnson & Johnson Vision has recently launched a new spherical contact lens, ACUVUE<sup>®</sup> OASYS with Transitions<sup>TM</sup>, that has photochromic properties. The purpose of this study is to evaluate the performance of the lens when fit as monovision in a presbyopic population who habitually wear monovision correction.

## 1.1. Name and Descriptions of Investigational Products

Test Lens: Over-labeled ACUVUE® OASYS with Transitions™.

## 1.2. Intended Use of Investigational Products

The study lenses are spherical lenses intended to correct refractive ametropia (myopia or hyperopia) in subjects who may have 1.00 D or less of refractive astigmatism. The lenses are intended to be used as a 2-week, reusable, daily wear lens. The lenses require use of a care system to clean and disinfect the lenses.

## 1.3. Summary of Findings from Nonclinical Studies

See the ACUVUE® OASYS with Transitions<sup>TM</sup> package insert in APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT).

## 1.4. Summary of Known Risks and Benefits to Human Subjects

See the ACUVUE® OASYS with Transitions<sup>TM</sup> package insert in APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT).

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

Refer to the ACUVUE® OASYS with Transitions $^{TM}$  package insert in APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT).

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

This study is an evaluation of the visual performance and subjective response of ACUVUE® OASYS with Transitions<sup>TM</sup> fit as monovision.

#### 2.2. Endpoints

The study endpoints will be the subjective CLUE Vision scores and logMAR visual acuity. Additional endpoints will be quantitative contrast sensitivity function (qCSF) measured at site 1036.

#### **Primary Endpoint**

• logMAR visual acuity scores, and CLUE vision scores

## Secondary Endpoint

N/A

#### Other Observations

• qCSF (Site 1036 only)

## 2.3. Hypotheses

The following primary hypotheses will be tested throughout this investigation.

## Primary Hypotheses:

- 1. After 10 to 14 days of wear, the distance, binocular, high luminance, high contrast visual acuity score for the Test lens will be statistically better than +0.01 logMAR.
- 2. After 10 to 14 days of wear, the intermediate, binocular, high luminance, high contrast visual acuity score for the Test lens will be statistically better than +0.17 logMAR.
- 3. After 10 to 14 days of wear, the near, binocular, high luminance, high contrast visual acuity score for the Test lens will be statistically better than +0.17 logMAR.
- 4. After the first 10 to 14 days of wear, the PRO CLUE vision scores for the Test lens will be statistically better than 32 CLUE points. This will be recorded by the subject using the CLUE Follow-up Questionnaire from Visit 2.

If all the primary hypotheses are met, the following secondary hypotheses will be tested.

## Secondary Hypotheses:

The PRO CLUE vision scores after the second 10 to 14 days wear cycle (Visit 4) will be statistically better than the score after the first 10 to 14 days wear cycle (Visit 2). This will be recorded using the CLUE Follow-up Questionnaire.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

Healthy male and female subjects who are habitual soft contact lens wearers will be recruited. Subjects will be at least 40 years of age and not older than 70 years of age. They will be myopic or hyperopic and have presbyopia.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all the following criteria to be enrolled in the study:

Inclusion Criteria after Screening:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.

- 2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. The subject must be between 40 and 70 years of age at the time of screening.
- 4. Subjects must own a wearable pair of spectacles if required for their distance vision.
- 5. The subject must be an adapted monovision soft contact lens wearer in both eyes (i.e., worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month of more duration).

#### Inclusion Criteria after Baseline:

- 6. The subject's distance spherical equivalent refraction must be in the range of +3.50 D to -4.00 D in each eye.
- 7. The subject's refractive cylinder must be  $\leq 1.00$  D in each eye.
- 8. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
- 9. The subject must have best corrected distance visual acuity of 20/20<sup>-3</sup> or better in each eye.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria after Screening:

- 1. Currently Pregnant or lactating.
- 2. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g., hepatitis, tuberculosis).
- 3. Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, oral phenothiazines (e.g., Haldol, Mellaril, Thorazine, Elavil, Pamelor, Compazine), systemic steroids.
- 4. Any previous, or planned, ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, dacryocystorhinostomy, etc.).
- 5. Use of any ocular medication, with the exception of rewetting drops.
- 6. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
- 7. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
- 8. Any known hypersensitivity or allergic reaction to OPTI-FREE® Puremoist® care cleaning solution, non-preserved rewetting drop solution or sodium fluorescein.
- 9. History of herpetic keratitis.
- 10. Entropion, ectropion, chalazia, glaucoma, history of recurrent corneal erosions.
- 11. A history of amblyopia, strabismus or binocular vision abnormality

Exclusion Criteria after Baseline

- 12. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
- 13. Any ocular infection or inflammation.
- 14. Any ocular abnormality that may interfere with contact lens wear.
- 15. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.

## 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

## 4. STUDY DESIGN AND RATIONALE

## 4.1. Description of Study Design

The clinical study is a single-ARM, single-masked, clinical trial. The mask will be a partial mask in that the lenses will be over-labeled and the specific brand of the contact lens will not be disclosed to the subject however the subject will be aware of the photochromic properties of the contact lens. There is one study treatment with two wearing cycles. A total of approximately 80 eligible subjects will be targeted to complete the study. The test article in the first wearing cycle will be dispensed for 12±2 days and at the follow-up the final lens measurements will occur. Subjects will complete a 7±3 days washout and then return for the second wearing cycle. New lenses with same power of the final pair from Visit 1 will be dispensed and the above sequence repeated. The lens in the second wearing cycle will not be optimized.

#### 4.2. Study Design Rationale

The study is intended to evaluate the initial performance, of a photochromic lens fit as monovision, in terms of the subjective response and visual acuity, after a period of lens dispensing. The single-ARM study is used as the performance will be measured against historical performance measures used in previous multifocal contact lens studies. A washout period and lens re-dispensing was used to evaluate the reproducibility and repeatability of the subjective vision response.

#### 4.3. Enrollment Target and Study Duration

A total of 80 subjects (48 myopes and 32 Hyperopes) are targeted to complete the study. The study will last approximately 3-5 months.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

The study lenses will be worn in a bilateral fashion using a single-arm design with 1 lens type and 2 wearing cycles.

## 5.2. Masking

This is a single-masked study with the subjects being masked. The lenses from different wearing cycles will be over-labeled using different letters so that the subjects don't know for sure the lenses are identical.

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken, the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

## 5.3. Procedures for Maintaining and Breaking the Masking

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- 1. Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule/randomization scheme to obtain the test article assignment for that subject prior to dispensing
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme if applicable.
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section.

## 6. STUDY INTERVENTION

## 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Test |
|---|---|
| Name | ACUVUE® OASYS with Transitions™ |
| Manufacturer | Johnson & Johnson® Vision, Inc. |
| Lens Material | senofilcon A |
| Nominal Base Curve | 8.4 mm |
| Nominal Diameter | 14.0 mm |
| Nominal Distance | +6.00 D to |
| Powers (D) | -4.00 D in 0.25 D steps |
| Nominal Cylinder | None |
| Powers (D) and Axes | |
| Nominal ADD Powers (D) | None |
| Water Content | 38% |
| Center Thickness | 0.085 mm |
| | (-3.00 D) |
| Oxygen Permeability<br>(Dk) | 121.0 |
| Wear Schedule in | Daily Wear Reusable |
| Current Study | VETTER YEARS ■ 10 NEW THEOGRAPH AND AND CONTROL BOOM |
| Replacement Frequency | Two Weeks |
| Packaging Form (vial, blister, etc.) | Blister |

# 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Single-Use Preservative-<br>three options may be supp | \$2.50 miles 100 | ions (any of these |
|---|---|---|---|
| Solution | Eye-Cept® Rewetting | ScleralFil® Preservative Free Saline Solution | LacriPure Saline |
| Name/Description | Drops | | Solution |

| Single-Use Preservative-Free Rewetting Solution three options may be supplied) | | | tions (any of these |
|---|---|---|---|
| Manufacturer | Optics Laboratory | B&L | Menicon |
| Preservative | Non-Preserved | Non-preserved | Non-preserved |

| | Solution |
|---|---|
| Solution<br>Name/Description | OPTI-FREE® Puremoist®<br>Multipurpose Disinfecting<br>Solution |
| Manufacturer | Alcon Laboratories |
| Preservative | Myristamidopropyl<br>dimethylamine 0.0005%<br>polyquaternium-1 0.001% |

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subject meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

## 6.4. Packaging and Labeling

The test articles will be packaged in blisters, as the primary packaging. The test article will be over-labeled to mask the subject to the identity of the lens. The test articles will be in investigational cartons sealed with a tamper evident seal, commercial cartons, or in plastic bags as the secondary packaging form. The sample study label is shown below:



## 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures and stored out of direct sunlight at the clinical site. Test articles must be kept under secure conditions.

CR-6349 v5.0 JJVC CONFIDENTIAL

## **6.6.** Collection and Storage of Samples

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return to JJV.

## 6.7. Accountability of Test Articles

JJV will provide the Investigator with sufficient quantities of study article and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test article must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits
- 2. What was returned to the Investigator unused
- 3. The number and reason for unplanned replacements

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to the Sponsor.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor immediately.

Site Instructions for Test Article Receipt and Test Article Accountability for additional information

# 7. STUDY EVALUATIONS

# 7.1. Time and Event Schedule

Table 3: Time and Events

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 |
|---------------------|------------|-------------|-----------|-----------|
| | Screening, | Treatment 1 | Baseline | Treatment |
| | Baseline, | Follow-up | Treatment | 2 Follow- |
| | Treatment | 7±3 Day | 2 Fitting | up |
| | 1 Fitting | Wash-out | | |
| Time Point | Day 0 | Day 12±2 | Day 7±3 | Day 12±2 |
| | | from V1 | from V2 | from V3 |
| Estimated Visit | 2.5 hours | 1.5 hour | 2.0 hour | 1.5 hour |
| Duration | | | | |
| Statement of | | | | |
| Informed Consent | X | | | |
| Demographics | X | | | |
| Medical | | | | |
| History/Concomitant | | | | |
| Medications | X | | | |
| Adverse Events and | | | | |
| Concomitant | | | | |
| Medications Review | | X | X | X |
| Compliance | | X | | X |
| Habitual Contact | | | | |
| Lens Information | X | | | |
| Contact Lens | | | | |
| History | X | | | |
| Wear Time and | | | | |
| Comfortable Wear | | | | |
| Time with lenses | X | X | | X |
| Screening | | | | |
| Inclusion/Exclusion | | | | |
| Criteria | X | | | |
| Subject Reported | | | | |
| Ocular Symptoms | X | X | X | X |
| Baseline PRO | | | | |
| (CLUE and MRD) | | | | |
| Questionnaires | X | | | |
| CLDEQ-8 | | | | |
| Questionnaire | X | X | | X |
| Baseline PRO | X | | X | |

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 |
|---|---|---|---|---|
| | Screening, | Treatment 1 | Baseline | Treatment |
| | Baseline, | Follow-up | Treatment | 2 Follow- |
| | Treatment | 7±3 Day | 2 Fitting | up |
| | 1 Fitting | Wash-out | | <b>.</b> . |
| Time Point | Day 0 | Day 12±2 | Day 7±3 | Day 12±2 |
| A CONTROL OF CASE OF CASE | 0.000.00 | from V1 | from V2 | from V3 |
| Estimated Visit | 2.5 hours | 1.5 hour | 2.0 hour | 1.5 hour |
| Duration | SERVICE SERVICES NERVOS | Shakini inganisani | | |
| (CLUE) | | | | - |
| Questionnaire | | | | |
| Distance and Near | | | | |
| Entrance Visual | | | | |
| Acuity | x | X | X | x |
| Lens Removal | | | x (if | |
| Lens Kemovai | X | X | applicable) | X |
| Keratometry | X | | | 3 |
| Subjective | | | | |
| Refraction and | | | | |
| Distance Visual | | | | |
| Acuity | X | | | |
| Near ADD | | | | |
| Determination | X | | | A |
| Ocular Dominance | X | | | |
| ADD Refinement | X | | 8 | |
| Near Visual Acuity | X | | | |
| Biomicroscopy | X | X | X | X |
| Baseline Inclusion/ | | | | |
| Exclusion Criteria | X | | | |
| Continuance | | | X | |
| Lens Selection | X | | X | |
| Lens Insertion | X | | X | |
| 10 Minute Settling | X | | X | |
| Visual Satisfaction / | | | | |
| Subjective | | | | |
| Acceptance | X | X | X | Х |
| Study Lens Distance | | | | |
| and Near Visual | | | | |
| Acuity | X | X | X | Х |
| Distance Over | | | | |
| Refraction and | | | | |
| Visual Acuity | X | X | X | r. |
| Lens Fit | | | | |
| Assessment | X | X | X | X |

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 |
|---------------------|------------|-------------|-----------|-----------|
| | Screening, | Treatment 1 | Baseline | Treatment |
| | Baseline, | Follow-up | Treatment | 2 Follow- |
| | Treatment | 7±3 Day | 2 Fitting | up |
| | 1 Fitting | Wash-out | | |
| Time Point | Day 0 | Day 12±2 | Day 7±3 | Day 12±2 |
| | | from V1 | from V2 | from V3 |
| Estimated Visit | 2.5 hours | 1.5 hour | 2.0 hour | 1.5 hour |
| Duration | | | | |
| Binocular Over | | | | |
| Refraction | | X | | X |
| Visual Performance | | X | | X |
| qCSF (Site 1036 | | | | |
| only) | X | X | | X |
| Modifications | X | | 2 | - |
| Post-Fit PRO | | | | |
| (MRD) | | | | |
| Questionnaire | X | | X | |
| Follow-up PRO | | | | |
| (CLUE and MRD) | | | | |
| Questionnaires | | X | | X |
| Distance and Near | | | | |
| Exit Visual Acuity | X | X | X | |
| Dispensing Criteria | X | | X | |
| Instructions | X | X | X | 2 |
| Schedule Next Visit | X | X | X | |
| Wash-out | | X | | |
| Final Evaluation | | | | X |

# 7.2. Detailed Study Procedures

## VISIT 1

Subjects must report to the visit wearing their habitual contact lenses to accurately assess baseline PRO (CLUE) performance. If the subject is not wearing their lenses they must be rescheduled.

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the |

| | | consent form. Note: The subject must be provided a signed copy of this document. |
|---|---|---|
| 1.2 | Demographics | Record the subject's age, gender, race and ethnicity. |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. |
| 1.4 | Habitual Lenses | Questions regarding the subject's habitual lens type and parameters. |
| 1.5 | Contact Lens History | Record the subject's correction type (i.e. monovision, multifocal, sphere with readers, etc.). |
| 1.6 | Wear time and<br>Comfortable Wear<br>time with Habitual<br>lenses | Record the subjects wear time and comfortable wear time with their habitual contact lenses. |
| 1.7 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. |

| į. | | Visit 1: Baseline | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.8 | Baseline PRO<br>(CLUE and MRD)<br>and CLDEQ-8<br>Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of their habitual lenses using the PRO (CLUE and MRD) questions. | |
| 1.9 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 1.10 | Entrance Visual<br>Acuity | Distance and near Snellen visual acuity will be measured for each eye with the subject's habitual contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | |
| 1.11 | Binocular Contrast<br>Sensitivity (CS)<br>Measurement (Site<br>1036 only) | Measure the subject's Binocular CS at 4M, distance. The measurement is made using the attached work aid. See section 4 to set the trial number (set to 25) and section 5 to execute the test. | Appendix<br>G |
| 1.12 | Lens Removal | Have the subject remove their habitual lenses and store in an approved storage solution. | |

| 1.13 | Keratometry | Keratometry will be performed OD and OS | |
|---|---|---|---|
| 1.15 | 1 Teracomou y | and the steep and flat dioptric power and | |
| | | corresponding meridians recorded. | |
| 1.14 | Subjective Refraction | An optimal, binocular balanced distance | |
| | and Distance Visual | sphero-cylindrical refraction will be | |
| | Acuity | performed. Record the refraction and distance | |
| | | visual acuity to the nearest letter. | |
| | | The same and the same street. | |
| | | Note: Best distance visual acuity with sphero- | |
| | | cylindrical refraction must be at least 20/20 <sup>-3</sup> | |
| | | in each eye for the subject to be eligible in the | |
| | | study. | |
| 1.15 | Near ADD | The near reading addition will be determined | |
| | Determination | using the binocular crossed cylinder technique | |
| | | (BCC) at 40 cm followed by optimization in a | |
| | | trial frame in step 1.16 below. | |
| 1.16 | Ocular Dominance | Determine the distance ocular dominance with | Appendix F |
| | | the best distance correction in place using a | |
| | | +1.00-blur test. If the results are equivocal use | |
| | | the sighting dominance test to determine the | |
| | | dominant eye used for the study. | |
| 1.17 | ADD Refinement | Place the BCC result in the trial frame and | |
| | | refine the near prescription with trial lenses (or | |
| | | flippers) under binocular conditions. | |
| 1.18 | Near Visual Acuity | Using the ETDRS 2000 Series Chart 1 or 2 | |
| | | near card placed at 40 cm. Record the near | |
| 1.10 | D' ' | visual acuity OD, OS and OU at 40 cm. | |
| 1.19 | Biomicroscopy | FDA Slit Lamp Classification Scale will be | |
| | | used to grade the findings and determine | |
| | | eligibility. | |
| | | For the conjunctival redness 0.5 | |
| | | unit increments will be used in the grading. | |
| | | Corneal Staining Assessment will | |
| | | be graded in 1.0 increments. | |
| | | If any of these slit lamp findings are Grade 3 | |
| | | or higher, the subject will be discontinued. If | |
| | | discontinued a final examination must be | |
| | | completed. | |
| | | r | |
| | | If the clearance of the fluorescein needs to be | |
| | | expedited, preservative-free rewetting drops or | |
| | | saline may be instilled. | |
| 1.20 | Eligibility after | All responses to Inclusion Criteria questions | |
| | Baseline | must be answered "yes" and all responses to | |
| | | Exclusion Criteria questions must be answered | |

| "no" for the subject to be considered eligible. |
|--------------------------------------------------|
| If so, proceed to lens fitting. If not, complete |
| the final evaluation and discharge the subject. |

| SF. | Visit 1: Treatment 1 Lens Fitting | | |
|---|---|---|---|
| Step | Procedure | Details | 30 |
| 1.21 | Lens Selection | Select the monovision lens pair based on the spherical equivalent of the distance refraction for the dominant eye and the spherical equivalent of the distance refraction plus the near ADD for the non-dominant eye. Record the Test lens parameters (power and lot number). | |
| 1.22 | Lens Insertion | Subjects will insert the lenses themselves. If the lens is uncomfortable, inspect for damage and remove, reinsert or replace as necessary. Damaged lenses will be stored in labeled vial with sterile saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. Complete the Quality Product Complaint form. | |
| 1.23 | Lens Settling | Allow the study lenses to settle for a minimum of 10 minutes. | |
| 1.24 | Determine Visual<br>Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look down a hallway or out of a window for distance vision assessments, and for them to read a book, magazine or similar for near vision. | |
| 1.25 | Study Lens Distance<br>and Near Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. Note: Use the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm to measure the Near visual acuity | |
| 1.26 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 1.27 | Subjective Lens Fit<br>Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and | |

| | | tightness (push-up test). |
|---|---|---|
| | | <ul> <li>The subject should not proceed to wear the lenses if any of the following is observed:</li> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> <li>If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form.</li> </ul> |
| 1.28 | Modifications | If the subject reports unsatisfactory vision or is unable to obtain 20/30 distance visual acuity OU with the lenses, then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and based upon their findings on the measured visual acuity and/or over- refraction the investigator may make a modification. Up to two attempts at modification are permitted if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Allow at least 10 minutes of settling time between each lens modification attempted. If modifications are required steps 1.21-1.27 will be repeated for each modification. |
| 1.29 | PRO (MRD) Post-Fit<br>Questionnaire | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO (MRD) questionnaire. |
| 1.30 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |

| 1.31 | Dispensing Criteria | Note: The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. The lenses will be dispensed for 10-14 days. • Distance Snellen acuity equal to or better than 20/30 OU • Subject must indicate that the vision is acceptable. • Subject must indicate that the comfort of the lenses is acceptable. |
|---|---|---|
| | | • Lenses must have an acceptable general lens fit. |
| 1.32 | Patient Instructions | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>OPTI-FREE® Puremoist® solution will be used in a rub regime to disinfect and store the lenses each night in the lens case provided.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>A patient instruction booklet will be provided.</li> <li>Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline and returned to the Sponsor.</li> </ul> |
| 1.33 | Schedule | The subject will be scheduled to return for |

| Follow-up | their follow-up appointment in 12±2 days. |
|---|---|
| | Note: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

## VISIT 2

The subjects must present to Visit 2 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| Visit 2: Treatment 1 Follow-up | | |
|---|---|---|
| Step | Procedure | Details |
| 2.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 2.2 | Wear Time | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 2.3 | Compliance | Record the subject's compliance with wearing the study lenses. Note: Subjects must have worn lenses for at least 6 hours per day To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. |
| 2.4 | PRO (CLUE and<br>MRD) and CLDEQ-8<br>Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO (CLUE and MRD) questionnaire. |
| 2.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire |
| 2.6 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. |
| 2.7 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 2.8 | Visual Performance<br>Distance (4M)<br>Intermediate (64 cm) | Visual performance will be recorded OD, OS, and OU for the following: Distance, Bright Illuminance |

| | Near (40 cm) | High and Low Contrast ETDRS Charts 4M- HC#1, HC#2, HC#3 and LC#1, LC#2, LC#3 Near, Bright Illuminance Reduced Guillon-Poling Charts Intermediate (64 cm) High Contrast and Low Contrast Near (40 cm) High Contrast and Low Contrast | |
|---|---|---|---|
| | | Distance, Dim Illuminance (with <u>Distance</u> goggles) High Contrast ETDRS Charts 4M-HC#4, HC#5, HC#6 | |
| | | Near, Dim Illuminance (with <u>Near goggles</u> ) Reduced Guillon-Poling charts High Contrast Intermediate (64 cm) and Near | |
| | | (40 cm). Note: • The room illuminance must be | |
| | | between 7.3 and 7.9 EV (394-597 lux). • Distance, HC-1 Chart luminance | |
| | | Acceptable Range 10.5-10.7 EV (181-208 cd/m²). • Guillon-Poling, Near Chart Luminance Acceptable Range 10.8-11.1 EV (223-274 cd/m²). | |
| | | Do not use the Mesopic filter for Dim<br>luminance (Dim luminance will be<br>simulated by using the goggles) | |
| 2.9 | Binocular Contrast<br>Sensitivity (CS)<br>Measurement (Site<br>1036 only) | Measure the subject's Binocular CS at 4M, distance. The measurement is made using the attached work aid. See section 4 to set the trial number (set to 25) and section 5 to execute the test. | Appendix<br>G |
| 2.10 | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. Note: No lens changes are allowed based on the over-refraction. | Appendix<br>D |
| 2.11 | Lens Fit Assessment: | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). | |
| | | The subject should not proceed to wear the | |

| lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze |
|---|
| clear cornea) in any gaze |
| - presence of odge lift |
| • presence of edge lift |
| • presence of unacceptable movement |
| (excessive or insufficient) in all three |
| movement categories (primary gaze, |
| upgaze, and push-up). |
| If either lens is deemed unacceptable, the |
| subject will be discontinued from the study. |
| Remove the lenses, perform a slit-lamp |
| evaluation, and complete the Final Evaluation |
| form. |
| 2.12 Lens Removal Have the subject remove the study lenses and |
| store in saline in a labeled glass vial. |
| <b>Note:</b> Lenses do not need to be stored in a |
| refrigerator. |
| 2.13 Biomicroscopy Perform biomicroscopy OD and OS. Slit Lamp |
| Classification Scales will be used to grade the |
| findings. |
| For the conjunctival redness 0.5 |
| unit increments will be used in the grading. |
| Corneal Staining Assessment will |
| be graded in 1.0 increments. |
| If the clearance of the fluorescein needs to be |
| expedited, preservative-free rewetting drops or |
| saline may be instilled. |
| 2.14 Exit Visual Acuity Distance and near Snellen visual acuity will be |
| measured for each eye with the subject's |
| habitual correction lenses in place. |
| For near measures use the ETDRS 2000 Series |
| Chart 1 or 2. The acuity will be recorded to |
| the nearest letter OD, OS and OU. |
| 2.15 Subject Instructions Subjects will complete a wash out period of |
| 7±3 days. |
| Instruct the subjects they can wear their |
| habitual contacts or glasses during the washout |
| period. |
| 2.16 Schedule Next Visit The subject will be scheduled to return for |
| their next visit in 4-10 days. |

## VISIT 3

Subjects must report to the visit wearing their habitual contact lenses to accurately assess baseline PRO (CLUE) performance. If the subject is not wearing their lenses they must be rescheduled.

| Visit 3: Baseline | | |
|---|---|---|
| Step | Procedure | Details |
| 3.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 3.2 | Baseline PRO<br>(CLUE<br>Questionnaire) | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of their habitual lenses using the PRO (CLUE) questions. |
| 3.3 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 3.4 | Entrance Visual<br>Acuity | Record the distance and near Snellen visual acuity with the subjects' habitual correction in place (OD, OS, and OU) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. Note: Use the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm to measure the Near visual acuity. |
| 3.5 | Lens Removal | Have the subject remove their habitual lenses and store in an approved storage solution. |
| 3.6 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. For the conjunctival redness 0.5 unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. If any of these slit lamp findings are Grade 3 |
| | | or higher, the subject will be discontinued. If discontinued a final examination must be completed. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or |

| | | saline may be instilled. |
|---|---|---|
| 3.7 | Continuance | Determine whether the subject is eligible to continue in the study based on the examination findings. |

| Visit 3: Treatment 2 Lens Fitting | | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 3.8 | Lens Selection | Select the monovision power based on the | 1.8 |
| 0.5-47-45-0.0 | A TO SO SOMETHIS TO SO SO AND AN ADD SO AND A SOCIETY | lens power dispensed at Visit 1. Record the | |
| | | Test lens parameters (power and lot number). | |
| 3.9 | Lens Insertion | Subjects will insert the lenses themselves. If | |
| | | the lens is uncomfortable, inspect for damage | |
| | | and remove, reinsert or replace as necessary. | |
| | | VIII. 1011 1111 1111 1111 1111 1111 1111 | |
| | | Damaged lenses will be stored in labeled vial | |
| | | with sterile saline, and clearly differentiated | |
| | | from the other worn lenses that will be | |
| | | shipped back to the Sponsor. Complete the | |
| 5 | | Quality Product Complaint form. | |
| 3.10 | Lens Settling | Allow the study lenses to settle for a | |
| | | minimum of 10 minutes. | |
| 3.11 | Determine Visual | Determine if the subject's vision is acceptable | |
| | Satisfaction | with the lenses. Allow the subject to look | |
| | | down a hallway or out of a window for | |
| | | distance vision assessments, and for them to | |
| | | read a book, magazine or similar for near | |
| | | vision. | |
| | | <i>Note:</i> If the subject's vision is unacceptable | |
| | | the subject will be discontinued. Complete the | |
| | | final evaluation. (No Modifications allowed) | |
| 3.12 | Distance and Near | Measure the distance and near visual acuity | |
| | Entrance Visual | OD, OS and OU. Record the results. | |
| | Acuity | | |
| | | For near measures use the ETDRS 2000 | |
| | | Series Chart 1 or 2. The acuity will be | |
| | | recorded to the nearest letter OD, OS and OU. | |
| 3.13 | Distance Over- | Perform a distance over-refraction OD and OS | |
| | Refraction and | using loose lenses outside of the phoropter | |
| | Distance Visual | under ambient room illumination. The | |
| | Acuity | distance over-refraction may also be refined | |
| | | under binocular conditions. Record the | |
| | | results. The results of the distance over- | |
| | | refraction may also be checked for the impact | |
| | | on near vision under monocular and/or | |
| | | binocular conditions. | |
| 3.14 | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. | |
|---|---|---|--|
| | | An unacceptable fit is deemed by one of the following criteria: • limbal exposure at primary gaze or with extreme eye movement; • edge lift; • excessive movement in primary and up gaze; or • insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up. | |
| | | If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. | |
| 3.15 | PRO (MRD) Post-Fit<br>Questionnaire | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO (MRD) questionnaire. | |
| 3.16 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. Note: The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. | |
| 3.17 | Dispensing Criteria | <ul> <li>The lenses will be dispensed for 12±2 days.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> </ul> | |

| 3.18 | Patient Instructions | <ul> <li>The lenses will be worn on a daily wear basis.</li> <li>OPTI-FREE® Puremoist® solution will be used in a rub regime to disinfect and store the lenses each night in the lens case provided.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>Subjects will be instructed to bring their habitual contacts or spectacles to the next visit.</li> </ul> |
|---|---|---|
| 3.19 | Schedule<br>Follow up | Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline and returned to the Sponsor. The subject will be scheduled to return for their follow up appointment in 12+2 day. |
| | Follow-up | Note: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

# VISIT 4

The subjects must present to Visit 4 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 4: Treatment 2 Follow-up 1 | |
|---|---|---|
| Step | Procedure | Details |
| 4.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 4.2 | Wear Time | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 4.3 | Compliance | Record the subject's compliance with wearing the study lenses. Note: Subjects must have worn lenses for at least 6 hours per day To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. |
| 4.4 | PRO (CLUE and<br>MRD) and CLDEQ-8<br>Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO (CLUE and MRD) questionnaire. |
| 4.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire |
| 4.6 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. |
| 4.7 | Distance and Near<br>Entrance Visual<br>Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the |
| 4.8 | Visual Performance<br>Distance (4M)<br>Intermediate (64 cm)<br>Near (40 cm) | nearest letter OD, OS and OU. Visual performance will be recorded OD, OS, and OU for the following: Distance, Bright Illuminance High and Low Contrast ETDRS Charts 4M- HC#1, HC#2, HC#3 and LC#1, LC#2, LC#3 |

| | T | | · |
|---|---|---|---|
| | | Near, Bright Illuminance Reduced Guillon-Poling Charts Intermediate (64 cm) High Contrast and Low Contrast Near (40 cm) High Contrast and Low Contrast | |
| | | Distance, Dim Illuminance (with <u>Distance</u> goggles) High Contrast ETDRS Charts 4M-HC#4, HC#5, HC#6 Near, Dim Illuminance (with <u>Near</u> goggles) Reduced Guillon-Poling charts High Contrast Intermediate (64 cm) and Near (40 cm). | |
| | | <ul> <li>Note:</li> <li>The room illuminance must be between 7.3 and 7.9 EV (394-597 lux).</li> <li>Distance, HC-1 Chart luminance Acceptable Range 10.5-10.7 EV (181-208 cd/m²).</li> <li>Guillon-Poling, Near Chart</li> </ul> | |
| | | Luminance Acceptable Range 10.8- | |
| | | 11.1 EV (223-274 cd/m <sup>2</sup> ). | |
| | | <ul> <li>Do not use the Mesopic filter for Dim<br/>luminance (Dim luminance will be</li> </ul> | |
| | | simulated by using the goggles) | |
| 4.9 | Binocular Contrast<br>Sensitivity (CS)<br>Measurement (Site<br>1036 only) | Measure the subject's Binocular CS at 4M, distance. The measurement is made using the attached work aid. See section 4 to set the trial number (set to 25) and section 5 to execute the test. | Appendix<br>G |
| 4.10 | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. Note: No lens changes are allowed based on the over-refraction. | Appendix<br>D |
| 4.11 | Lens Fit Assessment: | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). | |
| | | The subject should not proceed to wear the lenses if any of the following is observed: | |
| | | • presence of limbal exposure (appearance of clear cornea) in any gaze | |

| | | presence of edge lift presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. |
|---|---|---|
| 4.12 | Lens Removal | Have the subject remove the study lenses and store in saline in a labeled glass vial. Note: Lenses do not need to be stored in a refrigerator. |
| 4.13 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. For the conjunctival redness 0.5 unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |

# FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Distance Subjective<br>Sphero-cylindrical<br>Refraction and<br>Distance Exit Visual<br>Acuity | An optimal, binocular balanced distance sphero-cylindrical refraction will be performed. Record the refraction and distance visual acuity to the nearest letter. |
| F.2 | Subject Disposition | Indicate if the subject completed the study successfully. If subject discontinued from the study indicate the reason. |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected at a minimum:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate
- Date and time of the visit and all procedures completed at the unscheduled visit
- Review of adverse event and concomitant medications
- Documentation of any test article dispensed or collected from the subject, if applicable
- Slit lamp findings (using the Slit Lamp Classification Scale)

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pre-treatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| U.1 | Chief Complaints | Record the subject's chief complaints for reasons for the unscheduled visit |
| U.2 | Adverse Events and<br>Concomitant Medications<br>Review | Review the subject's concomitant medications and record any changes from the previous study visit. |
| U.3 | Subject Reported Ocular<br>Symptoms | Subjects will respond to a verbal open-<br>ended symptoms questionnaire. |
| U.4 | Entrance VA | Record the entrance distance and near visual acuity (OD, OS and OU) to the nearest letter. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| U.5 | Subjective Sphero-<br>cylindrical Refraction | An optimal, binocular balanced distance sphero-cylindrical refraction will be performed. |

| | Unscheduled Visit | | |
|---|---|---|---|
| | Record the refraction and distance visual | | |
| | | acuity to the nearest letter. | |
| U.6 | Biomicroscopy | FDA Slit Lamp Classification Scale will be | F |
| *************************************** | | used to grade the findings and determine | |
| | | eligibility. | |
| | | | e <del></del> |
| | | For the conjunctival redness 0.5 | |
| | | unit increments will be used in the grading. | |
| | | Corneal Staining Assessment | |
| | | will be graded in 1.0 increments. | |
| | | 00 g 110 | |
| | | If the clearance of the fluorescein needs to | |
| | | be expedited, preservative-free rewetting | |
| | | drops or saline may be instilled. | |
| U.7 | Lens Dispensing | Additional study lenses may be dispensed | |
| · · · | Dens Dispensing | when required. | |
| U.8 | Lens Fit Assessment: | Evaluate and grade lens centration, primary | |
| 0.0 | | gaze movement, upgaze movement and | |
| | | tightness (push-up test). | |
| | | against (Fact of 1999). | |
| | | The subject should not proceed to wear the | |
| | | lenses if any of the following is observed: | |
| | | presence of limbal exposure (appearance) | |
| | | of clear cornea) in any gaze | |
| | | presence of edge lift | |
| | | <ul> <li>presence of unacceptable movement</li> </ul> | |
| | | (excessive or insufficient) in all three | |
| | | movement categories (primary gaze, | |
| | | upgaze, and push-up). | |
| | | If either lens is deemed unacceptable, the | |
| | | subject will be discontinued from the study. | |
| | | Remove the lenses, perform a slit-lamp | |
| | | evaluation, and complete the Final | |
| | | Evaluation form. | |
| U.9 | Exit Visual Acuity | Record the subject's exit distance and near | |
| 0.7 | DAIL VISUAL MEURLY | visual acuity (OD, OS and OU) to the | |
| | | nearest letter. | |
| | | nearest letter. | |
| | | For near measures use the ETDRS 2000 | |
| | | Series Chart 1 or 2. The acuity will be | |
| | | recorded to the nearest letter OD, OS and | |
| | | OU. | |
| i. | | 00. | |

## 7.4. Laboratory Procedures

Not Applicable.

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

## 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent
- they are eligible
- completed all study visits

# 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period
- Subject withdrawal of consent
- Subject not compliant to protocol
- Subject lost to follow-up
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant)
- Subject develops significant or serious adverse events causing discontinuation of study lens wear
- Subjects who have experienced a Corneal Infiltrative Event (CIE)
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)
- Subject missed two consecutive study visits
- Subject not compliant with study lens wear schedule
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study
- Record the spherocylindrical refraction with best corrected distance visual acuity
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 6.7.
- Collect all unused test article(s) from the subject

An additional subject may be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications and therapies are medications or therapies that contraindicate contact lens wear. See the Exclusion criteria for specific details.

## 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Major protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked, and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJV reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJV, it is determined that it would be unwise to continue at the clinical site.

JJV (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated, as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

# 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)"
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site
- Lens replacements that occur due to drops/fall-outs
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness)
- Who received the complaint
- Study number
- Clinical site information (contact name, site ID, telephone number)
- Lot number(s)
- Unique Subject Identifier(s)
- Indication of who first observed complaint (site personnel or subject)
- OD/OS indication, along with whether the lens was inserted
- Any related AE number if applicable
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.)
- Eye Care Provider objective (slit lamp) findings if applicable
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.

*Note 1* to entry: This definition includes events related to the investigational medical device or the comparator.

*Note 2* to entry: This definition includes events related to the procedures involved.

*Note 3* to entry: For users or other persons, this definition is restricted to events related to investigational medical devices."<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study
- 2. Was present prior to the study but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event

**Serious Adverse Event (SAE)** – An SAE is any untoward medical occurrence that:

- Results in death
- Is life threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity (e.g., a sight threatening event, a significant persistent or permanent change, impairment, damage, or disruption to the subject's body)
- Is a congenital anomaly/birth defect
- Requires intervention to prevent permanent damage (the use of the test article
  resulting in a condition which requires medical or surgical intervention to preclude
  permanent impairment of the body structure or a body function). Important medical
  events that may not result in death, be life-threatening, or require hospitalization may
  be considered an SAE when, based upon appropriate medical judgment, they may

jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in the above definition

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – Those events that are usually symptomatic and warrant discontinuation (temporary or permanent) of the test article (excluding Serious Adverse Events).

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of >2 Lines of BSCVA
- Other Grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation >2 weeks

**Non-Significant Adverse Events** – Those conditions that are usually asymptomatic and usually do not warrant discontinuation (temporary or permanent) of the test article. However, the Investigator may choose to treat as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis

- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation <2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device.

*Note 1* to entry: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

*Note 2* to entry: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device."

Unanticipated Adverse Device Effect (UADE) – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

# 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1)
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; unlikely related; possibly related; related see definition in Section 13.2.1)
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild; moderate; severe for all events see definition in Section 13.2.2)
- Outcome not recovered or not resolved; recovering or resolving; recovered or resolved with sequelae; recovered or resolved; death related to adverse event; unknown
- Actions Taken none; temporarily discontinued; permanently discontinued; other.

## 13.2.1. Causality Assessment

**Causality Assessment** – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely

- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge.

## 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities.

# 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begins when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

• Adverse event (diagnosis not symptom)

- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.)
- Date the clinical site was notified
- Date and time of onset
- Date and time of resolution
- Adverse event classification, severity, and relationship to test articles, as applicable
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements
- Any referral to another health care provider if needed
- Outcome, ocular damage (if any)
- Likely etiology
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the test article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

# 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

## 13.4.1. Reporting Adverse Events to Sponsor

# **Serious/Significant Adverse Events**

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations

## **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

## **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

## 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

## 13.4.3. Event of Special Interest

None.

## 13.5. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. At the Investigator's discretion, the study participant may be followed by the Investigator through delivery. However, this data will not be collected as part of the clinical study database. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

#### 14.1. General Considerations

All data summaries and statistical analyses will be performed using the Statistical Analysis System (SAS) software Version 9.4 (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (Descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation [SD], median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

Summaries will be presented by study lens type and will be performed separately by completion status (Safety Population or Per-Protocol Population). All analyses will be conducted on per-protocol population (see Section 14.3).

## 14.2. Sample Size Justification

A total of 80 subjects (48 myopes and 32 hyperopes) are targeted to complete the study.

Using the POWER procedure in SAS 9.4, below is the summary of sample size required based on the different assumptions of the true LogMAR visual acuity and CLUE scores. The sample size was calculated for the non-inferiority tests (using 0.05 as the margin) with at least 90% of statistical power and 2-sided type I error of 0.05. Assuming the true LogMAR visual acuity is between 0.00 to 0.05 (distance) or 0.08 to 0.12 (near), and true CLUE vision score is between 38 to 42 points.

## • Binocular LogMAR visual acuity (distance)

| | Estimated Standard | | Actual |
|------------|--------------------|----------------------|--------|
| True Value | Deviation | # of subjects needed | Power |
| 0.00 | 0.12 | 18 | 0.915 |
| 0.02 | 0.12 | 26 | 0.904 |
| 0.05 | 0.12 | 63 | 0.902 |

# • Binocular LogMAR visual acuity (intermediate and near)

| | Estimated Standard | | Actual |
|------------|--------------------|----------------------|--------|
| True Value | Deviation | # of subjects needed | Power |
| 0.08 | 0.12 | 21 | 0.905 |
| 0.10 | 0.12 | 33 | 0.901 |
| 0.12 | 0.12 | 63 | 0.902 |

## • CLUE vision score

| | Estimated Standard | | Actual |
|------------|--------------------|----------------------|--------|
| True Value | Deviation | # of subjects needed | Power |
| 38 | 17 | 87 | 0.902 |
| 40 | 17 | 50 | 0.903 |
| 42 | 17 | 33 | 0.906 |

## 14.3. Analysis Populations

## **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

## **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the Per-Protocol Population set will be documented in a memo to file.

## **Intent-to-Treat (ITT) Population:**

All subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

## 14.4. Level of Statistical Significance

All planned analysis for this study will be conducted with an overall type I error rate of 5%.

## 14.5. Primary Analysis

Primary efficacy analysis:

Binocular, high luminance, high contrast logMAR visual acuity will be analyzed using a linear mixed model. The model will include the experimental design factors: distance (distance/intermediate/near) and time point (2 week or 4 week) as fixed effects; and site and subject nested in site as random effects. Other baseline characteristics known to be important such as age, gender, subject group (myope/hyperope), and/or ADD power will be included as fixed covariates when appropriate. The covariance between residual errors from the same subject at the same time point across distances will be selected based on the finite-sample corrected Akaike's Information Criterion. Covariance structures considered will include: Homogenous Compound Symmetry (CS), Heterogeneous Compound Symmetry (CSH), and Unstructured covariance structure (UN). The structure that returns the lowest Akaike Information Criteria Corrected (AICC) will be selected as the structure that best fit the data. Heterogeneous models across study populations and/or distance will be considered using a log-likelihood ratio test.

Comparisons will be carried out using 95% confidence intervals (CIs) constructed of Least-square means (LSM) from the linear mixed models. Statistical superiority will be concluded if the upper limit of the confidence intervals of the Test lens is below +0.10 logMAR for distance, and below +0.17 logMAR for intermediate and near.

## **CLUE Vision**

Overall quality of vision scores will be analyzed using a linear mixed model adjusting for baseline values as fixed covariates. The model will include the experimental design factors: time point (2 week or 4 week) as the fixed effect; and site and subject nested in site as random effects. Other baseline characteristics known to be important such as age, gender, subject group (myope/hyperope), and/or ADD power will be included as fixed covariates when appropriate. The covariance between residual errors from the same subject across lens wearing periods/time point will be selected based on the finite-sample corrected Akaike's Information Criterion. Covariance structures considered may include: Homogenous compound symmetry (CS) and Unstructured covariance structure (UN). The structure that returns the lowest Akaike Information Criteria Corrected (AICC) will be selected as the structure that best fit the data.

# Primary Hypothesis:

Comparisons will be carried out using 95% confidence intervals constructed of least-square means (LSM) from the linear mixed models of CLUE vision scores at the end of first wearing cycle (2 week). Statistically superiority will be concluded if the lower limit of the confidence intervals of the test lens are greater than 32 points.

#### Secondary Hypothesis:

Comparisons between the wearing cycles (2 week vs 4 week) will be carried out using 95% confidence intervals constructed of least-square means (LSM) differences (4 week - 2 week) from the linear mixed model. The superiority will be established if the lower confidence limit is above 0.

In all models, the Kenward and Roger method<sup>7</sup> will be used for the calculation of the denominator of degrees of freedom.

## 14.6. Secondary Analysis

Secondary efficacy analysis: See section 14.5

## 14.7. Other Exploratory Analyses

Not Applicable.

## 14.8. Interim Analysis

Not Applicable.

# 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis will be conducted using multiple imputation methods if the proportion of subject dropout is greater than the 15%. The SAS/STAT procedures PROC MI and PROC MIANALYZE will be utilized with a parametric regression method used to make at least 5 imputations.

# 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

## 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system (Bioclinica). An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJV database manager and sent to JJV for analysis.

External Date Sources for this study include: Not Applicable.

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives

will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.<sup>1</sup>

# 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable.

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

## 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJV must be contacted and notified in writing within 24 hours.

## 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJV. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJV will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

## 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJV may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJV and for inspection by local and regulatory authorities.

#### 17. MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent amendments, and regulatory requirements are maintained
- Ensuring the rights and wellbeing of subjects are protected
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel
- Ensuring that protocol deviations are documented with corrective action plans, as applicable
- Ensuring that the clinical site has sufficient test article and supplies
- Clarifying questions regarding the study
- Resolving study issues or problems that may arise

• Reviewing of study records and source documentation verification in accordance with the monitoring plan.

#### 18. ETHICAL AND REGULATORY ASPECTS

# 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

## 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

## 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol and, if applicable, amendments
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information) and amendments
- Sponsor-approved subject recruitment materials
- Information on compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB)
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects
- Any other documents that the IEC/IRB requests to fulfill its obligation.

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, amendments (if any), the informed consent form, applicable recruiting materials,

and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure amendments or new edition(s)
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB.

For protocol amendments that increase subject risk, the amendment and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

Each subject must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will

be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>5</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

#### 18.5. Privacy of Personal Data

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations. The Sponsor ensures that the personal data will be:

- processed fairly and lawfully
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes
- adequate, relevant, and not excessive in relation to said purposes
- accurate and, where necessary, kept current.

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable

steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJV.

## 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJV management representative prior to study initiation.

JJV reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study
- Scheduling a study visit outside the subject's acceptable visit range

JJV reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution
- Case Report Form signature
- Completion of any follow-up action items

# 21. PUBLICATION

This study will be registered on ClinicalTrials.gov by the Sponsor.

#### 22. REFERENCES

- 1. ISO 14155:2011: Clinical Investigation of Medical Devices for Human Subjects Good Clinical Practice. Available at: https://www.iso.org/standard/4557.html
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP). Available at: http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. Available at: https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- 4. United States (US) Code of Federal Regulations (CFR). Available at: https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR
- 5. *Health Information Portability and Accountability Act (HIPAA)*. Available at: https://www.hhs.gov/hipaa/for-professionals/privacy/index.html
- Keselman HJ, Algina J, Kowalchuk RK, Wolfinger RD. A Comparison of Two Approaches for Selecting Covariance Structures in the Analysis of Repeated Measures. Communications in Statistics—Simulation and Computation. 1998;27:591-604.
- 7. Kenward MG, Roger JH. Small Sample Inference for Fixed Effects from Restricted Maximum Likelihood. *Biometrics*. 1997;53:983–997.

# APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)







5

PRO SPECIFICATIO


4 Final 2019-06-18




JJVC CONFIDENTIAL

Protocol 6349



12








16













Protocol 6349


Protocol 6349



# APPENDIX B: PATIENT INSTRUCTION GUIDE

Patient Instruction Guide will be provided separately.

# APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

IMPORTANT: Please read carefully and keep this information for future use.

This Package Insert and Fitting Instruction Guide is intended for the Eye Care Professional, but should be made available to patients upon request.

The Eye Care Professional should provide the patient with the appropriate instructions that pertain to the patient's prescribed lenses. Copies are available for download at www.acuvue.com.



ACUVUE® OASYS Contact Lenses with Transitions™

senofilcon A Soft (hydrophilic) Contact Lenses with UV Blocker and Photochromic Additive for Daily Wear Only



# SYMBOLS KEY

The following symbols may appear on the label or packaging:

| SYMBOL | DEFINITION |
|---|---|
| <b>△</b> □i | Caution, Consult Instructions for Use |
| <b></b> | Manufacturer |
| سا | Date of Manufacture |
| $\square$ | Use by Date (Expiration Date) |
| LOT | Batch Code |
| STERILE | Sterilized Using Steam Heat |
| C€ <sub>0086</sub> | Quality System Certification Symbol |
| UV BLOCKING | UV Blocking |
| 0 | Fee Paid for Waste Management |
| Ŷ | Lens Orientation Correct |
| $\stackrel{\vee}{\times}$ | Lens Orientation Incorrect (Lens Inside Out) |
| EC REP | Authorized Representative in the European Community |
| 8 | Do Not Use if Package is Damaged |
| * | Store Away from Direct Sunlight |

 $\label{thm:com-guides} \mbox{ Visit www.acuvue.com/guides for additional information about symbols.}$ 

#### DESCRIPTION

ACUVUE® OASYS with Transitions™ are soft (hydrophilic) contact lenses available as spherical lenses. The lenses are made of a silicone hydrogel material (senofilcon A) containing an internal wetting agent, and UV absorbing monomers.

A combination of the benzotriazole UV absorbing monomer and the naphthopyran monomer (photochromic additive) is used to block UV radiation.

The transmittance characteristics for these lenses are less than 1% in the UVB range of 280 nm to 315 nm and less than 10% in the UVA range of 316 nm to 380 nm for the entire power range.

Additionally, the photochromic additive absorbs visible light in the range from 380 nm to 780 nm to a minimum 84% transmittance in the inactivated (closed) state. The activated (open) state dynamically absorbs visible light dependent on the lens thickness and the level of UV and high energy visible (HEV) radiation to a minimum of 23% transmittance.

#### **Lens Properties**

The physical/optical properties of the lens are:

Specific Gravity (calculated): 0.98 - 1.12

• Refractive Index: 1.42

Visible Light Transmission – 84% minimum

inactivated:

Visible Light Transmission – 23% minimum

activated (calculated):

Surface Character: Hydrophilic

Water Content: 38%

Oxygen Permeability (Dk):

#### VALUE METHOD

103 x 10-11 (cm²/sec) Fatt (boundary corrected, (ml O $_z$ /ml x mm Hg) at 35°C edge corrected)

122 x 10<sup>-11</sup> (cm²/sec) Fatt (boundary corrected, (ml O<sub>x</sub>/ml x mm Hg) at 35°C non-edge corrected)

## Lens Parameters Ranges:

Diameter (DIA): 12.0 mm to 15.0 mm
 Center Thickness: Varies with power
 Base Curve (BC): 7.85 mm to 10.00 mm
 Spherical Power (D): -20.00D to +20.00D

## **AVAILABLE LENS PARAMETERS**

ACUVUE® OASYS with Transitions™ contact lenses are hemispherical shells of the following dimensions:

Diameter (DIA): 14.0 mm

Center Thickness: 0.085 mm to 0.217 mm

(varies with power)

**Base Curve (BC):** 8.4 mm, 8.8 mm **Powers (D):** -12.00D to +8.00D

#### TRANSMITTANCE CURVES

ACUVUE® OASYS with Transitions™ contact lens vs. 24 yr. old human cornea vs. 25 yr. old human crystalline lens.



\*The data was obtained from measurements taken through the central 2 mm x 7.5 mm portion for the thinnest marketed lens (-0.25D lens, 0.085 mm center thickness).

\*Leman, S., Radiant Energy and the Eye, MacMillan, New York, 1980, p. 58, figure 2-21.

\*Waxler, M., Hitchins, V.M., Optical Radiation and Visual Health, CRC Press, Boca Raton,

Florida, 1986, p. 19, figure 5.

The data was obtained from measurements taken through the central 6 mm portion for the thinnest marketed lines (-0.25D lens, 0.085 mm center thickness). The method for measuring the transmittance in the activated state is based on visible range 380 nm to 780 nm utilizing a spectrophotometer and an activation source. **Note:** There is no impact to the level of UV blocking in the activated state compared to the inactivated state.

#### **ACTIONS**

In its hydrated state, the contact lens, when placed on the cornea, acts as a refracting medium to focus light rays on the retina.

A combination of the benzotriazole UV absorbing monomer and the naphthopyran monomer (photochromic additive) is used to block UV radiation.

The transmittance characteristics are less than 1% in the UVB range of 280 nm to 315 nm and less than 10% in the UVA range of 316 nm to 380 nm for the entire power range.

The photochromic additive dynamically absorbs visible light allowing for the attenuation of bright light. These lenses absorb visible light in the range from 380 nm to 780 nm to a minimum 84% transmittance in the inactivated (closed) photochromic state and to a minimum of 23% transmittance in the activated (open) photochromic state dependent on the lens thickness and the level of absorbed UV and high energy visible (HEV) radiation.

WARNING: UV absorbing contact lenses are NOT substitutes for protective UV absorbing eyewear, such as UV absorbing goggles or sunglasses because they do not completely cover the eye and surrounding area. The patient should continue to use UV absorbing eyewear as directed.

NOTE: Long-term exposure to UV radiation is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as environmental conditions (altitude, geography, cloud cover) and personal factors (extent and nature of outdoor activities). UV blocking contact lenses help provide protection against harmful UV radiation. However, clinical studies have not been done to demonstrate that wearing UV blocking contact lenses reduces the risk of developing cataracts or other eye disorders. The Eye Care Professional should be consulted for more information.

### INDICATIONS (USES)

ACUVUE® OASYS with Transitions™ contact lenses (spherical) are indicated for daily wear for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may have 1.00D or less of astigmatism.

These lenses are also indicated for the attenuation of bright light as they contain a photochromic additive which dynamically absorbs visible light.

These lenses contain a UV blocker to help protect against transmission of harmful UV radiation to the cornea and into the eye.

Eye Care Professionals may prescribe the lenses for frequent/ planned replacement wear with cleaning, disinfection and scheduled replacement (see REPLACEMENT SCHEDULE). When prescribed for frequent/planned replacement wear, the lenses may be disinfected using a chemical disinfection system only and should be discarded after the recommended wearing period as prescribed by the Eye Care Professional.

When the lenses are worn in a frequent/planned replacement modality, they are intended to be worn for up to 2 weeks (14 days).

#### CONTRAINDICATIONS (REASONS NOT TO USE)

**DO NOT USE** these lenses when any of the following conditions exist:

- Acute or subacute inflammation or infection of the anterior chamber of the eye.
- Any eye disease, injury, or abnormality that affects the cornea, conjunctiva, or eyelids.
- · Severe insufficiency of lacrimal secretion (dry eye).
- Corneal hypoesthesia (reduced corneal sensitivity).
- Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses.
- Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses or use of contact lens solutions.
- Ocular irritation due to allergic reactions which may be caused by use of contact lens solutions (e.g. cleaning and disinfecting solutions, rewetting drops, etc.) that contain chemicals or preservatives (such as mercury, Thimerosal, etc.) to which some people may develop an allergic response.
- Any active corneal infection (bacterial, fungal, protozoal, or viral)
- · If eyes become red or irritated.

#### **WARNINGS**

Patients should be advised of the following warnings pertaining to contact lens wear.

EYE PROBLEMS, INCLUDING CORNEAL ULCERS, CAN DEVELOP RAPIDLY AND LEAD TO LOSS OF VISION. IF THE PATIENT EXPERIENCES:

- · Eye Discomfort,
- · Excessive Tearing,
- · Vision Changes,
- · Loss of Vision,
- · Eye Redness, or
- · Other Eye Problems,

# THE PATIENT SHOULD BE INSTRUCTED TO IMMEDIATELY REMOVE THE LENSES AND PROMPTLY CONTACT THE EYE CARE PROFESSIONAL.

- Patients should be instructed not to wear their lenses while sleeping. Clinical studies have shown that when daily wear users wear their lenses overnight (outside the intended indication), the risk of ulcerative keratitis is greater than among those who do not wear them overnight.<sup>4</sup>
- Studies have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than nonsmokers.
- Problems with contact lenses or lens care products could result in serious injury to the eye. Patients should be cautioned that proper use and care of contact lenses and lens care products, including lens cases, are essential for the safe use of these products.
- The overall risk of ulcerative keratitis may be reduced by carefully following directions for lens care, including cleaning the lens case.

<sup>4</sup> New England Journal of Medicine, September 21, 1989; 321 (12), pp. 773-783.

8

#### Specific Instructions for Use and Warnings:

#### Water Activity

#### Instruction for Use

Do not expose contact lenses to water while wearing them.

#### WARNING:

Water can harbor microorganisms that can lead to severe infection, vision loss, or blindness. If lenses have been submersed in water when participating in water sports or swimming in pools, hot tubs, lakes, or oceans, the patient should be instructed to discard them and replace them with a new pair. The Eye Care Professional should be consulted for recommendations regarding wearing lenses during any activity involving water.

#### Soaking and Storing Your Lenses

#### Instruction for Use

Use only fresh multi-purpose (contact lens disinfecting) solution each time the lenses are soaked (stored).

#### **WARNING**

Do not reuse or "top-off" old solution left in the lens case since solution reuse reduces effective lens disinfection and could lead to severe infection, vision loss, or blindness.

"Topping-Off" is the addition of fresh solution to solution that has been sitting in the case.

## • Discard Date on Multi-Purpose Solution Bottle Instructions for Use

- -Discard any remaining solution after the recommended time period indicated on the bottle of multi-purpose solution used for disinfecting and soaking the contact lanses
- -The discard date refers to the time that the patient can safely use the contact lens care product after the bottle has been opened. It is not the same as the expiration date, which is the last date that the product is still effective before it is opened.

#### WARNING:

Using multi-purpose solution beyond the discard date could result in contamination of the solution and can lead to severe infection, vision loss, or blindness.

- -To avoid contamination, DO NOT touch tip of container to any surface. Replace cap after using.
- -To avoid contaminating the solution, DO NOT transfer to other bottles or containers.

#### • Rub and Rinse Time

#### Instruction for Use

To adequately disinfect the lenses, the patient should rub and rinse the lenses according to the recommended lens rubbing and rinsing times in the labeling of the multipurpose solution.

#### WARNING:

- -Rub and rinse lenses for the recommended amount of time to help prevent serious eye infections.
- -Never use water, saline solution, or rewetting drops to disinfect the lenses. These solutions will not disinfect the lenses. Not using the recommended disinfectant can lead to severe infection, vision loss, or blindness.

#### Lens Case Care

#### Instructions for Use

- -Empty and clean contact lens cases with digital rubbing using fresh, sterile disinfecting solution/contact lens cleaner. Never use water. Cleaning should be followed by rinsing with fresh, sterile disinfecting solutions (never use water) and wiping the lens cases with fresh, clean tissue is recommended. Never air-dry or recap the lens case lids after use without any additional cleaning methods. If air-drying, be sure that no residual solution remains in the case before allowing it to air-dry.
- Replace the lens case according to the directions provided by the Eye Care Professional or the manufacturer's labeling that accompanies the case.
- -Contact lens cases can be a source of bacterial growth.

#### WARNING:

Do not store lenses or rinse lens cases with water or any non-sterile solution. Only fresh multi-purpose solution should be used to prevent contamination of the lenses or lens case. Use of non-sterile solution can lead to severe infection, vision loss, or blindness.

#### **PRECAUTIONS**

#### Special Precautions for Eye Care Professionals:

 Due to the small number of patients enrolled in clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated in significant numbers. Consequently, when selecting an appropriate lens design and parameters, the Eye Care Professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, wettability, central and peripheral thickness, and optic zone diameter.

The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore, the continuing ocular health of the patient and lens performance on the eye should be carefully monitored by the prescribing Eye Care Professional.

- Patients who wear these lenses to correct presbyopia using monovision may not achieve the best corrected visual acuity for either far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.
- Eye Care Professionals should instruct the patient to remove lenses immediately if the eyes become red or irritated.

- Eye Care Professionals should inform the patient that there is no data available on the safety driving performance with ACUVUE® OASYS with Transitions™ contact lenses for individuals age 50 and older who may have lens opacities.
- Eye Care Professionals should instruct the patient to always have a functional pair of spectacles with a current prescription available to use if the patient becomes unable to wear contact lenses, or in circumstances where contact lens wear is not advised.

Eye Care Professionals should carefully instruct patients about the following care regimen and safety precautions.

#### **Handling Precautions:**

- DO NOT use if the sterile blister package is opened or damaged.
- Always wash and rinse hands before handling lenses. It is best to put on lenses before putting on makeup.
- Carefully follow the handling, insertion, removal, cleaning, disinfecting, storing and wearing instructions in the PATIENT INSTRUCTION GUIDE for these lenses and those prescribed by the Eye Care Professional.
- Never use tweezers or other tools to remove lenses from the lens container. Slide the lens up the side of the bowl until it is free of the container.

## **Lens Wearing Precautions:**

- If the lens sticks (stops moving) on the eye, follow the recommended directions in "Care for a Sticking (Non-Moving) Lens." The lens should move freely on the eye for the continued health of the eye. If non-movement of the lens continues, the patient should be instructed to immediately consult his or her Eye Care Professional.
- Never wear lenses beyond the period recommended by the Eye Care Professional.

- The patient should be advised to never allow anyone else to wear their lenses. Sharing lenses greatly increases the chance of eye infections.
- If aerosol products, such as hairspray, are used while wearing lenses, exercise caution and keep eyes closed until the spray has settled.
- Avoid all harmful or irritating vapors and fumes while wearing lenses.
- Be aware that wearing a darkened ACUVUE® OASYS with Transitions™ lens on only one eye is not recommended because it may cause disturbances in the patient's ability to accurately judge depth and the motion of objects. It may also create a cosmetic concern. Therefore, unilateral vision correction is not recommended for ACUVUE® OASYS with Transitions™ contact lenses; it is recommended that a 0.00D photochromic lens be worn on the other eye in this instance.
- Be aware that ACUVUE® OASYS with Transitions™
  contact lenses are not intended for use as protection
  against artificial light sources, such as sun lamps, lasers,
  etc.
- The patient should be advised to never stare directly at the sun or at an eclipse with or without ACUVUE® OASYS with Transitions™ contact lenses.
- The patient should be advised to never rinse the lenses in water from the tap. Tap water contains many impurities that can contaminate or damage the lenses and may lead to eye infection or injury.

#### **Lens Care Precautions:**

- Different solutions cannot always be used together and not all solutions are safe for use with all lenses. Use only recommended solutions.
- Never use solutions recommended for conventional hard contact lenses only.

- Always use fresh, unexpired lens care solutions and lenses. Always follow directions in the package inserts for the use of contact lens solutions.
- Do not change solution without consulting with the Eye Care Professional.
- Sterile unpreserved solutions, when used, should be discarded after the time specified in the directions.
- Do not use saliva or anything other than the recommended solutions for lubricating or wetting lenses.
- Always keep the lenses completely immersed in the recommended storage solution when the lenses are not being worn (stored). Prolonged periods of drying (e.g. exposing the lens to air for 30 minutes or more) will reduce the ability of the lens surface to return to a wettable state. If the lens surface does become dried out, discard the lens and use a new one.
- Always store worn ACUVUE® OASYS with Transitions™ contact lenses in the lens case and out of direct sunlight.

#### Other Topics to Discuss with Patients:

- Always contact the Eye Care Professional before using any medicine in the eyes.
- Certain medications, such as antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers and those for motion sickness may cause dryness of the eye, increased lens awareness, or blurred vision. Should such conditions exist, proper remedial measures should be prescribed.
- Oral contraceptive users could develop visual changes or changes in lens tolerance when using contact lenses. Patients should be cautioned accordingly.
- Do not change lens type (e.g. brand name, etc.) or parameters (e.g. diameter, base curve, lens power, etc.) without consulting the Eye Care Professional.

- Instruct patients to always confirm the lens parameters printed on the multi-pack and on the individual lens package match their prescription. If there is a mismatch, the patient should not use the product.
- As with any contact lens, follow-up visits are necessary to assure the continuing health of the patient's eyes. The patient should be instructed as to a recommended followup schedule.
- Always store individual unopened blisters of ACUVUE® OASYS with Transitions™ out of direct sunlight.

# Who Should Know That the Patient Is Wearing Contact Lenses?

- Patients should inform all doctors (Health Care Professionals) about being a contact lens wearer.
- Patients should always inform their employer of being a contact lens wearer. Some jobs may require use of eye protection equipment or may require that the patient not wear contact lenses.

#### ADVERSE REACTIONS

# The patient should be informed that the following problems may occur when wearing contact lenses:

- · The eye may burn, sting, and/or itch.
- There may be less comfort than when the lens was first placed on the eye.
- There may be a feeling of something in the eye (foreign body, scratched area).
- There may be the potential for some temporary impairment due to peripheral infiltrates, peripheral corneal ulcers, or corneal erosion. There may be the potential for other physiological observations, such as local or generalized edema, corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis and conjunctivitis, some of which are clinically acceptable in low amounts.
- There may be excessive watering, unusual eye secretions, or redness of the eye.
- Poor visual acuity, blurred vision, rainbows, or halos around objects, photophobia, or dry eyes may also occur if the lenses are worn continuously or for too long a time.
- The patient should be instructed to conduct a simple 3-part self-examination at least once a day. They should ask themselves:
  - How do the lenses feel on my eyes?
  - How do my eyes look?
  - Have I noticed a change in my vision?

If the patient reports any problems, he or she should be instructed to IMMEDIATELY REMOVE THE LENS. If the problem or discomfort stops and the lens appears undamaged, the patient should clean and rinse the lens with a recommended contact lens care solution and reinsert the lens. If after reinserting the lens, the problem continues, the patient should discard the lens and place a new fresh lens on the eye.

If after inserting the new lens, the problem continues, the patient should be directed to IMMEDIATELY REMOVE THE LENS AND CONTACT HIS OR HER EYE CARE PROFESSIONAL.

The patient should be advised that when any of the above symptoms occur, a serious condition such as infection, corneal ulcer, neovascularization, or iritis may be present. He or she should be instructed to seek immediate professional identification of the problem and prompt treatment to avoid serious eye damage.

#### **GENERAL FITTING GUIDELINES**

#### A. Patient Selection

Patients selected to wear these lenses should be chosen based on:

- · Motivation to wear lenses
- · Ability to follow instructions regarding lens wear care
- · General health
- · Ability to adequately handle and care for the lenses
- · Ability to understand the risk and benefit of lens wear

Patients who do not meet the above criteria should not be provided with contact lenses.

## **B. Pre-Fitting Examination**

Initial evaluation of the patient should begin with a thorough case history to determine if there are any contraindications to contact lens wear. During the case history, the patient's visual needs and expectations should be determined as well as an assessment of their overall ocular, physical, and mental health.

Preceding the initial selection of trial contact lenses, a comprehensive ocular evaluation should be performed that includes, but is not limited to, the measurement of distance and near visual acuity, distance and near refractive prescription (including determining the preferred reading distance for presbyopes), baseline keratometry, and biomicroscopic evaluation.

Based on this evaluation, if it is determined that the patient is eligible to wear these lenses, the Eye Care Professional should proceed to the appropriate lens fitting instructions outlined

#### C. Initial Power Determination

A spectacle refraction should be performed to establish the patient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if the refraction is greater than  $\pm 4.00D$ .

17

#### D. Base Curve Selection (Trial Lens Fitting)

The following trial lens should be selected for the patient regardless of keratometry readings. However, corneal curvature measurements should be performed to establish the patient's baseline ocular status.

## • ACUVUE® OASYS with Transitions™: 8.4 mm/14.0 mm

The trial lens should be placed on each of the patient's eyes and evaluated after the patient has adjusted to the lenses.

#### 1 Criteria of a Properly Fit Lens

A properly fit lens will center and completely cover the cornea (i.e. no limbal exposure), have sufficient movement to provide tear exchange under the contact lens with the blink, and be comfortable. The lens should move freely when manipulated digitally with the lower lid, and then return to its properly centered position when released.

#### 2. Criteria of a Flat Fitting Lens

A flat fitting lens may exhibit one or more of the following characteristics: decentration, incomplete corneal coverage (i.e. limbal exposure), excessive movement with the blink, and/or edge standoff. If the lens is judged to be flat fitting, it should not be dispensed to the patient.

## 3. Criteria of a Steep Fitting Lens

A steep fitting lens may exhibit one or more of the following characteristics: insufficient movement with the blink, conjunctival indentation, and resistance when pushing the lens up digitally with the lower lid. If the lens is judged to be steep fitting, it should not be dispensed to the patient.

If the initial trial base curve is judged to be flat or steep fitting, the alternate base curve, if available, should be trial fit and evaluated after the patient has adjusted to the lens. The lens should move freely when manipulated digitally with the lower lid, and then return to a properly centered position when released.

## E. Final Lens Power (Spherical)

A spherical over-refraction should be performed to determine the final lens power after the lens fit is judged acceptable. The spherical over-refraction should be combined with the trial lens power to determine the final lens prescription. The patient should experience good visual acuity with the correct lens power unless there is excessive residual astigmatism.

| Example 1 | |
|----------------------------|--------|
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | -0.25D |
| Final lens power: | -2.25D |
| Example 2 | 3 |
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | +0.25D |
| Final lens power: | -1.75D |

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If the fit is acceptable, dispense the lenses and instruct the patient to return in one week for reassessment (see PATIENT MANAGEMENT section).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

## MONOVISION FITTING GUIDELINES

#### A. Patient Selection

## 1. Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. The amblyopic patient or the patient with significant astigmatism (greater than 1.00D) in one eye may not be a good candidate for monovision correction with these lenses.

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it should be determined by trial whether this patient can function adequately with monovision correction. Monovision contact lens wear may not be optimal for activities such as:

- Visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities, and
- Driving automobiles (e.g. driving at night). Patients who cannot pass their state driver's licensing requirements with monovision correction should be advised to not drive with this correction, OR may require that additional over-correction be prescribed.

#### 2. Patient Education

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with spectacles (multifocal, bifocal, trifocal, readers, progressives). Each patient should understand that monovision, as well as other presbyopic alternatives, can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments (e.g. reading a menu in a dimly lit restaurant, driving at night in rainy/foggy conditions, etc.). During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision, and straight ahead and upward gaze that monovision contact lenses provide.

#### **B. Eye Selection**

#### 1. Ocular Preference Determination Methods

Generally, the non-dominant eye is corrected for near vision. The following two methods for eye dominance can be used.

Method 1: Determine which eye is the "sighting eye."
Have the patient point to an object at the far end of the room. Cover one eye. If the patient is still pointing directly at the object, the eye being used is the dominant

(sighting) eye.

Method 2:

Determine which eye will accept the added power with the least reduction in vision while both eyes are open. Place a hand-held trial lens equal to +1.00D in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the +1.00D lens over the right or left eye, which is the non-dominant eye.

## 2. Other Eye Selection Methods

Other methods include the "Refractive Error Method" and the "Visual Demands Method."

#### Refractive Error Method:

For anisometropic correction, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.

#### Visual Demands Method:

Consider the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

Example: A secretary who places a copy to the left side of the desk will function best with the near lens on the

## C. Special Fitting Characteristics

#### 1. Unilateral Vision Correction

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens, whereas a bilateral myope would require corrective lenses on both eyes.

#### Examples

A presbyopic emmetropic patient who requires a +1.75D ADD would have a +1.75D lens on the near eye and the other eye left without correction.

A presbyopic patient requiring a +1.50D ADD who is -2.50D myopic in the right eye and -1.50D myopic in the left eye may have the right eye corrected for distance and the left uncorrected for near.

Note: Unilateral vision correction is not recommended for ACUVUE® OASYS with Transitions™ contact lenses. Having a darkened lens on only one eye may cause disturbances in the patient's ability to accurately judge depth and the motion of objects. It may also create a cosmetic concern. It is recommended that a 0.00D photochromic contact lens be worn on the other eye in this instance.

#### 2. Near ADD Determination

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

#### 3. Trial Lens Fitting

A trial fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the GENERAL FITTING GUIDELINES for base curve selection described in this Package Insert.

Case history and a standard clinical evaluation procedure should be used to determine the prognosis. Determine the distance correction and the near correction. Next determine the near ADD. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

Allow the lenses to settle for about 20 minutes with the correct power lenses in place. Walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernails. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tests are completed should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g. typewritten copy) at first and then graduate to newsprint and finally smaller type sizes.

After the patient's performance under the above conditions is completed, tests of visual acuity and reading ability under conditions of moderately dim illumination should be attempted.

An initial unfavorable response in the office, while indicative of a guarded prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

#### 4. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches, and a feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable, familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

#### **D. Other Suggestions**

The success of the monovision technique may be further improved by having the patient follow the suggestions below:

- Have a third photochromic contact lens (distance power) to use when critical distance viewing is needed.
- Have a third photochromic contact lens (near power) to use when critical near viewing is needed.
- Having supplemental spectacles to wear over the monovision contact lenses for specific visual tasks may improve the success of monovision correction. This is particularly applicable for those patients who cannot pass state driver's licensing requirements with monovision correction.
- Make use of proper illumination when carrying out visual tasks.

Monovision fitting success can be improved by the following suggestions:

- Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients.
- Emphasize the benefits of clear near vision, and straight ahead and upward gaze with monovision.

The decision to fit a patient with monovision correction is most appropriately left to the Eye Care Professional in conjunction with the patient after carefully considering the patient's needs.

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

## PATIENT MANAGEMENT

- Follow the accepted standard of care in fitting and following up with your patient.
- Schedule the appropriate follow-up examination.
- Preferably, at the follow-up visits, lenses should have been worn for at least six hours.
- Provide the patient with a copy of the Patient Instruction Guide for these lenses, which can be found at www.acuvue.com. REVIEW THESE INSTRUCTIONS WITH THE PATIENT SO THAT HE OR SHE CLEARLY UNDERSTANDS THE PRESCRIBED WEARING AND REPLACEMENT SCHEDULE (FREQUENT REPLACEMENT) AS WELL AS THE INFORMATION SPECIFIC TO WEARING PHOTOCHROMIC LENSES.
- Recommend an appropriate cleaning and disinfection system and provide the patient with instructions regarding proper lens care. Chemical or hydrogen peroxide disinfection is recommended.

## WEARING SCHEDULE

The wearing schedule should be determined by the Eye Care Professional. Regular checkups, as determined by the Eye Care Professional, are also extremely important.

Patients tend to over wear the lenses initially. The Eye Care Professional should emphasize the importance of adhering to the initial maximum wearing schedule. Maximum wearing time should be determined by the Eye Care Professional based upon the patient's physiological eye condition, because individual response to contact lenses varies.

Studies have not been completed to show that the lens is safe to wear while sleeping.

## REPLACEMENT SCHEDULE

The replacement schedule should be determined by the Eye Care Professional based upon the patient's history and their ocular examination, as well as the practitioner's experience and clinical judgment.

When prescribed for daily wear (frequent replacement), it is recommended that the lenses be discarded and replaced with a new lens every 2 weeks (14 days).

Once removed, it is recommended that the lens remains out of the eye for a period of rest of overnight or longer and be discarded in accordance with the prescribed replacement schedule.

## LENS CARE DIRECTIONS

For complete information concerning contact lens handling, care, cleaning, disinfecting and storage, refer to the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

The Eye Care Professional should review with the patient lens care directions for cleaning, disinfecting and storing, including both basic lens care information and specific instructions on the lens care regimen recommended for the patient.

### Care for a Sticking (Non-Moving) Lens

During removal, if the lens sticks to the eye, the patient should be instructed to apply a few drops of the recommended lubricating or rewetting solution directly to the eye and wait until the lens begins to move freely on the eye before removing it. If non-movement of the lens continues after a few minutes, the patient should **immediately** consult the Eye Care Professional.

#### **EMERGENCIES**

The patient should be informed that if chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the patient should: FLUSH EYES IMMEDIATELY WITH TAP WATER AND IMMEDIATELY CONTACT THE EYE CARE PROFESSIONAL OR VISIT A HOSPITAL EMERGENCY ROOM WITHOUT DELAY.

## **HOW SUPPLIED**

Each UV absorbing sterile lens is supplied in a foil-sealed plastic package containing borate buffered saline solution with methyl ether cellulose. The plastic package is marked with the following:

 ACUVUE® OASYS with Transitions™: base curve, power, diameter, lot number, and expiration date

## REPORTING OF ADVERSE REACTIONS

All serious adverse experiences and adverse reactions observed in patients wearing these lenses or experienced with the lenses should be reported to:

Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA Tel: 1-800-843-2020 www.acuvue.com

27

Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA Tel: 1-800-843-2020

www.acuvue.com



20407530

©Johnson & Johnson Vision Care, Inc. 2018 In Canada: Johnson & Johnson Vision Care, division of Johnson & Johnson, Inc. In USA: Johnson & Johnson Vision Care, Inc. Printed in USA Revision date: 11/2018

ACUVUE® OASYS is a trademark of Johnson & Johnson Vision Care, Inc.

Transitions™ and the Transitions logo are trademarks of Transitions Optical, Inc. used under license by TOL and JJVCI.

# APPENDIX D: BINOCULAR OVER REFRACTION

# Binocular Over-refraction Technique

- 1. Place trial frame on subject
- 2. Add +1.00 D sphere to OS
- 3. Add + 0.50DS OD and check VA
  - if VA remained unchanged or improved, repeat step 3
  - if VA decreased, add minus until best VA first achieved \*note: add minus for 0.5 seconds to avoid reflex accommodation.
- 4. Record VA
- 5. Change +1.00 D sphere to OD
- 6. Repeat steps 3 and 4

# APPENDIX E: PRESBYOPIC SYMPTOMS QUESTIONNAIRE

# **Presbyopic Symptoms Questionnaire**

- 1. Do you notice that you often have to hold things farther away so that you can read them?
- 2. Do you notice that you often have difficulty focusing on near objects (i.e., experiencing blurry vision when looking at things close-up)?
- 3. Do you often have headaches or eyestrain, or feel fatigued, when reading or conducting other near activities?
- 4. Do you often have difficulty reading small or fine prints, such as phone books, medicine bottles or package labels, etc.?
- 5. Do you often have difficulty reading under dim or low light?

# OCULAR DOMNANCE TEST

## +1.00 D LENS TEST

- Step 1 Place the subjects best sphero-cylindrical distance refraction in a trial frame.
- Step 2 Have the subject view a BVA line of letters.
- Step 3 With both eyes open alternate a +1.00 D trial lens between the right and left eye and ask the subject to indicate over which eye does the lens cause the line of letters to appear more blurred. The eye that the greatest blur is reported is the distance dominant eye. If the subject indicates that the amount of blur is about the same between the two eyes then record as neither eye dominant.

## SIGHTING OCULAR DOMINANCE

- Step 1 Ask the subject to extend both arms out and use his/her hands to form a triangle. The subject will be asked to keep both eyes open and look through the triangle at a small object on the wall (e.g., a light switch or doorknob).
- Step 2 Occlude the subject's left eye, then right eye. While alternating the occluder from the subject's eyes, ask the subject when they see the object.

If the subject sees the object when the left eye is covered, the subject is *right eye* dominant.

If the subject sees the object when the right eye is covered, the subject is *left eye* dominant.

If the subject sees the object with both eyes, the opening between the hands may be too large. Therefore, ask the subject to make a smaller opening and repeat the procedure.

## APPENDIX G: AST SENTIO CONTRAST SENSITIVITY TESTING

Work Aid: AST Sentio Contrast Sensitivity Testing

## **OBJECTIVE**

To provide instructions for capturing contrast sensitivity data using the AST Sentio Pro Instrument.

## DESCRIPTION

The AST Sentio is a vision testing system that consists of a monitor, internal computer, custom software, and remote control for registering user responses. The display, computer, and software are contained in one unit; the remote is separate. During testing, the monitor will show test patterns of varying sizes and contrasts. The particular pattern that is displayed during the test is determined by the custom software. During a test session, 25 or 50 triplets of test letters will be displayed, and the operator will record the patient's responses using the remote. After a test session is complete, the custom software will calculate the following.

Area under the log contrast sensitivity function from 1.5 cycles per degree to 18 cycles per degree output of a testing session. This metric is referred to as the AULCFS.

The highest spatial frequency at which a stimulus at full contrast is visible. This is equivalent to the intersection of the CSF curve and the X-axis. This metric is referred to as CFS Acuity.

## **MATERIALS**

AST Sentio Pro Monitor display with internal computer (see Figure 1). AST Sentio Remote (see Figure 1).





Figure 1: AST Sentio Pro Monitor (main unit) and Remote. The monitor has a USB port for data export. To start the remote, press the On/O button once. When the remote is on, to put the device into a hold mode, press the On/O button. The remote has a micro-USB port for charging.

## **SETUP**

The viewing distance for the AST Sentio Pro (ASP) instrument is 4 meters. This *cannot* be changed during the protocol.

Place the ASP so that no light sources create glare on the screen. Ensure no direct light sources are in the patient's field of view when the patient is facing the screen.

Plug the monitor into an AC 110V 50/60Hz grounded outlet. Do not use an extension cord. Ensure that the remote is charged. The remote has a micro-USB port for charging. When charging the remote, use a different AC outlet from the one that is being used for the monitor.

To start the remote, press the On/O button once. This will also start the main unit. When the remote is on, to put the device into a hold mode, press the On/O button.

Press [Settings] on the Main Screen to switch settings (see Figure 2).

Set the number of trials (either 25 or 50) using the [Number of Trials] slider in the Settings screen (see figure 2).



Figure 2: Main screen and settings screen

Using the [Show Info] button will display the following information Software revision (computer and remote).

Battery charge state (percentage of full charge).

Wi-Fi signal strength and name of Wi-Fi network.

Connection status to computer.

Connection status to monitor.

MAC address of computer adapter.

Percentage of storage space (hard drive) in computer.

## **TESTING**

Ensure that the remote is charged.

Ensure that the subject is positioned at the proper viewing distance (4 meters).

Ensure the subject's eyes, in primary gaze, are at 130 cm  $\pm$  10 cm from the ground.

Ensure that there is no glare on the screen or in the subject's field of view.

Instruct the subject as follows.

Inform the subject that they will be presented with letters of different sizes and contrast (faintness) on the monitor. These letters may not have a familiar appearance; they may be modified for testing purposes.

Inform the subject that they will be shown a short demonstration to familiarize them with the letters and procedure.

Inform the subject that they will encounter letters that they will not be able to identify or see and this is not an indication of poor visual performance. The purpose of the test is to find the limits of visual performance.

Inform the subject that if the subject is unsure about a letter, they should still respond. If this happens during the test, encourage the subject to respond.

Start the system by pressing the On/O button on the remote. The two screens in Figure 3 should be visible (one following the other).



Figure 3: After pressing the On/O button the system will power up and the Sentio remote will connect to the computer software. The screen on the left will be visible on the Sentio remote while the remote is attempting to connect. After the connection is made, the screen (Main Screen) will appear on the Sentio remote.

The demo mode can be accessed by pressing the "Demo" button on the main screen (see Figure 3). In the demo mode a screen as shown in Figure 4 will displayed on the Sentio remote. To advance to the next trial press the ">" symbol (see Figure 4). A total of 5 trials can be viewed in the demo mode. The system will return to the main screen once the last demo trial has been viewed. To stop the demo before the fifth trial, press the "stop" button (see Figure 4).



To start a test, press the ">" button on the main screen. This will advance to the setup screen on the Sentio Remote (see Figure 5).



Figure 5: Left image shows main screen; right image shows setup screen

Using the setup screen on the Sentio Remote, enter the subject ID (see protocol governing test).

Choose the appropriate eye (OS or OS) or both eyes (OU). See protocol governing test. Press the ">" button to start the test.

When the test is started, the monitor will show three letters with decreasing (left to right) visibility. The Sentio remote will show the correct identity of these letters. Be certain that the subject cannot see the Sentio remote screen.

Record the subject response as either correct (check mark) or incorrect (X). See Figure 6. Encourage the subject to name a letter; however, if the subject will not name a letter, record "no answer".

If the subject cannot see which letter is under consideration, or any letter, the test administrator can highlight the area containing the letter by pressing the prompt button (see Figure 6).

Press the ">" button to advance to the next trial. See Figure 6.



Figure 6: Sentio Remote screen in Test mode. The check box indicates a correct response (under letter D); the X indicates an incorrect response (under the letter R); and "no answer" indicates the subject would not offer a response (under the letter C). The prompt button is located at the top right under the number 01.

The "<" button acts as a back button and can be used if the test administrator incorrectly recorded a response. Note: in Figure 6, this button is not visible since it shows trial 1.

To abort the current test, press the "stop" button (next to the prompt button). A window will appear to confirm that the test is to be aborted.

After a set number of trials, pressing the ">" button will advance to the Results screen. See Figure 7.



Figure 7: results screen shown on Sentio remote. The green triangles denote a correct response, the red crosses denote an incorrect response, and the red slashes denote that no answer was given. The top of the screen displays the AULCSF and CSF acuity metrics.

Press the "Finish Test" button on the top right of the results screen (see Figure 7). After this is done a dialog box will appear (see Figure 8).



Figure 8: dialog box that will appear after pressing the "Finish Test" button on the results screen

To finish the test, press the "return to main" button in the dialog box (see Figure 8).

To start a new test with the same subject, press the "Same" button (see Figure 8).

To start a new test with a new subject, press the "New" button (see Figure 8).

## FOLLOWING A TEST

Exportation of Data

Press the "Return to Main" button. See 5.22.

All data are stored on the computer's hard drive and exportation of data may occur at any time. To export the data, insert a USB drive into the USB port on the front column of the cart.

At the main screen on the Sentio remote, click the export data button. You will be prompted with a dialog box asking to enter a password (see Figure 9). Enter a password (see protocol). After entering a password, press either "Export New", which will export the last data set, or press "Export All", which will export all subject data. Two files will be exported: a PDF and a JAVA file; each contains the data shown on the results screen.

## Continue Testing

Press either the "Same" or "New" buttons. See 5.23 and 5.24.

## Power Down

To turn the device off, press the On/O button on the Sentio remote. The monitor will count down for 10 seconds before powering down. If you wish to stop this, press the On/O button again; this will stop the device from powering down.

The device will power down if left inactive for some period of time. To restart the device, press the On/O button. Ongoing test results will be saved.

Do not unplug the device during testing; data for an ongoing test will not be saved.

## REFERENCES

AST Sentio Pro Instructions for Use. Software version 1.1. If U version 2016-08-07.

# APPENDIX H:

- LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS
- EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING
- DETERMINATION OF NEAR ADD
- NEAR logMAR VISUAL ACUITY MEASUREMENT PROCEDURE
- LENS FITTING CHARACTERISTICS
- SUBJECT REPORTED OCULAR SYMPTOMS
- DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS
- BIOMICROSCOPY SCALE
- KERATOMETRY
- DISTANCE AND NEAR VISUAL ACUITY EVALUATION
- ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE
- VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING

# LIMBAL AND CONJUNCTIVAL (BULBAR) REDNESS
















# EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING











## DETERMINATION OF NEAR ADDITION
























## NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE





Page 2 of 2

## LENS FITTING CHARACTERISTICS
















## SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS



# DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS



















## BIOMICROSCOPY SCALE















## KERATOMETRY PROCEDURE


## DISTANCE AND NEAR VISUAL ACUITY EVALUATION








## DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE







Page 3 of 3



## VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING



| Title: | Visual Acuity Chart Luminance and Room Illumination Testing |
|--------|-------------------------------------------------------------|





| Title: | Visual Acuity | Visual Acuity Chart Luminance and Room Illumination Testing | |
|---|---|---|---|
| -2 | | | |
| <del></del> | | | <del></del> |



| Title: | Vis | Visual Acuity Chart Luminance and Room Illumination Testing | |
|---|---|---|---|
| | 0.00 | | 201 |



## PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

CR-6349 Evaluation of A Marketed Silicone Hydrogel Spherical Lens Used for Monovision Correction of Presbyopia

Version and Date: 5.0 Amendment 4 03 September 2019

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155,<sup>1</sup> GCP and ICH guidelines,<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> United States (US) Code of Federal Regulations (CFR),<sup>4</sup> and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| | Signature | Date |
| | Name and Professional Position (Printed) | _ |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |